CLINICAL TRIAL: NCT00781391
Title: A Phase 3, Randomized, Double-Blind, Double-Dummy, Parallel Group, Multi-Center, Multi-National Study for Evaluation of Efficacy and Safety of Edoxaban (DU-176b) Versus Warfarin In Subjects With Atrial Fibrillation - Effective Anticoagulation With Factor Xa Next Generation in Atrial Fibrillation (ENGAGE - AF TIMI - 48)
Brief Title: Global Study to Assess the Safety and Effectiveness of Edoxaban (DU-176b) vs Standard Practice of Dosing With Warfarin in Patients With Atrial Fibrillation
Acronym: EngageAFTIMI48
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: The TIMI Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DU176b-C-U301
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Results first posted 2015-03-25 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2015-03

CONDITIONS: Stroke; Atrial Fibrillation; Embolism
Keywords: Systemic embolic events
MeSH Terms: conditions — Stroke; Atrial Fibrillation; Embolism | interventions — Warfarin; edoxaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Warfarin/placebo edoxaban (Active Comparator): Warfarin tablets plus placebo Edoxaban tablets
  Interventions: Drug: warfarin tablets; Drug: placebo edoxaban
- high dose edoxaban/placebo warfarin (Experimental): Edoxaban tablets (60mg) plus warfarin placebo tablets
  Interventions: Drug: Edoxaban tablets (high dose regimen-60mg); Drug: placebo warfarin
- low dose edoxaban/placebo warfarin (Experimental): Edoxaban tablets (30mg) plus warfarin placebo tablets
  Interventions: Drug: Edoxaban tablets (low dose regimen-30mg); Drug: placebo warfarin

INTERVENTIONS:
Drug: warfarin tablets — Warfarin tablets plus Edoxaban placebo tablets each taken once daily for 24 months
  Arms: Warfarin/placebo edoxaban
Drug: Edoxaban tablets (high dose regimen-60mg) — Edoxaban tablets plus warfarin placebo tablets each taken once daily for 24 months
  Arms: high dose edoxaban/placebo warfarin
Drug: Edoxaban tablets (low dose regimen-30mg) — Edoxaban tablets plus warfarin placebo tablets each taken once daily for 24 months
  Arms: low dose edoxaban/placebo warfarin
Drug: placebo warfarin — placebo warfarin
  Arms: high dose edoxaban/placebo warfarin; low dose edoxaban/placebo warfarin
Drug: placebo edoxaban — placebo edoxaban
  Arms: Warfarin/placebo edoxaban

SUMMARY:
This study is to demonstrate the safety and efficacy profile, in two different dose regimens of Edoxaban (DU-176b), (an investigational new drug being tested for the prevention of stroke/systemic embolic events (SEE)), in individuals with atrial fibrillation. Patients will be randomized to one of three treatment groups: High Dose Regimen, Low Dose Regimen, & Warfarin. The expected duration of the study is 24 months.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older; male or female.
* Able to provide written informed consent.
* History of documented AF within the prior 12 months
* A moderate to high risk of stroke, as defined by CHADS2 index score of at least 2

Exclusion Criteria:

* Transient atrial fibrillation secondary to other reversible disorders
* Subjects with moderate or severe mitral stenosis, unresected atrial myxoma, or a mechanical heart valve
* Subjects with any contraindication for anticoagulant agents;
* Subjects with conditions associated with high risk of bleeding or have known or suspected hereditary or acquired bleeding disorders
* Females of childbearing potential including the following:

  * Females with a history of tubal-ligation
  * Females less than 2 years post-menopausal

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21105 (Actual)
Dates: Start 2008-11; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1004):
- United States (311):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Gilbert, Arizona
  - Glendale, Arizona
  - Lake Havasu City, Arizona
  - Sierra Vista, Arizona
  - Tempe, Arizona
  - Tucson, Arizona
  - Harrisburg, Arkansas
  - Hot Springs, Arkansas
  - Little Rock, Arkansas
  - Alhambra, California
  - Anaheim, California
  - Burbank, California
  - Chula Vista, California
  - Encinitas, California
  - Fountain Valley, California
  - Glendale, California
  - Healdsburg, California
  - Lakewood, California
  - Long Beach, California
  - Los Alamitos, California
  - Los Angeles, California
  - Los Banos, California
  - Mather, California
  - Merced, California
  - Newport Beach, California
  - Oceanside, California
  - Pacific Palisades, California
  - Palm Springs, California
  - Pismo Beach, California
  - Redondo Beach, California
  - Sacramento, California
  - San Diego, California
  - Santa Rosa, California
  - Torrance, California
  - Ventura, California
  - Aurora, Colorado
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Englewood, Colorado
  - Greeley, Colorado
  - Bridgeport, Connecticut
  - Guilford, Connecticut
  - Hamden, Connecticut
  - Manchester, Connecticut
  - New Haven, Connecticut
  - North Haven, Connecticut
  - Shelton, Connecticut
  - Stamford, Connecticut
  - Trumbull, Connecticut
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - Aventura, Florida
  - Chipley, Florida
  - Clearwater, Florida
  - Daytona Beach, Florida
  - DeBary, Florida
  - Deerfield Beach, Florida
  - Delray Beach, Florida
  - Hialeah, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Jacksonville Beach, Florida
  - Jupiter, Florida
  - Leesburg, Florida
  - Melbourne, Florida
  - Miami, Florida
  - Naples, Florida
  - Orange Park, Florida
  - Orlando, Florida
  - Ormond Beach, Florida
  - Panama City, Florida
  - Pembroke Pines, Florida
  - Pensacola, Florida
  - Plantation, Florida
  - Port Charlotte, Florida
  - Rockledge, Florida
  - Saint Augustine, Florida
  - Sarasota, Florida
  - St. Petersburg, Florida
  - Stuart, Florida
  - Tamarac, Florida
  - Tampa, Florida
  - The Villages, Florida
  - Vero Beach, Florida
  - West Palm Beach, Florida
  - Athens, Georgia
  - Atlanta, Georgia
  - Conyers, Georgia
  - Covington, Georgia
  - Cumming, Georgia
  - Savannah, Georgia
  - Snellville, Georgia
  - Tucker, Georgia
  - Watkinsville, Georgia
  - Waycross, Georgia
  - Woodstock, Georgia
  - Honolulu, Hawaii
  - Boise, Idaho
  - Hayden Lake, Idaho
  - Bannockburn, Illinois
  - Belleville, Illinois
  - Chicago, Illinois
  - Elgin, Illinois
  - Joliet, Illinois
  - Libertyville, Illinois
  - Maywood, Illinois
  - Melrose Park, Illinois
  - Oak Lawn, Illinois
  - Springfield, Illinois
  - Winfield, Illinois
  - Bloomington, Indiana
  - Munster, Indiana
  - Ames, Iowa
  - Council Bluffs, Iowa
  - Iowa City, Iowa
  - Shell Rock, Iowa
  - Wichita, Kansas
  - Bowling Green, Kentucky
  - Campbellsville, Kentucky
  - Elizabethtown, Kentucky
  - Richmond, Kentucky
  - Marrero, Louisiana
  - West Monroe, Louisiana
  - Auburn, Maine
  - Biddeford, Maine
  - Baltimore, Maryland
  - Bel Air, Maryland
  - Bethesda, Maryland
  - Lexington Park, Maryland
  - Rockville, Maryland
  - Salisbury, Maryland
  - Towson, Maryland
  - Westminster, Maryland
  - Ayer, Massachusetts
  - Boston, Massachusetts
  - Concord, Massachusetts
  - East Bridgewater, Massachusetts
  - Haverhill, Massachusetts
  - Methuen, Massachusetts
  - Worcester, Massachusetts
  - Bay City, Michigan
  - Benzonia, Michigan
  - Chelsea, Michigan
  - Commerce, Michigan
  - Detroit, Michigan
  - Grand Rapids, Michigan
  - Interlochen, Michigan
  - Kalamazoo, Michigan
  - Lapeer, Michigan
  - Midland, Michigan
  - Rochester Hills, Michigan
  - Saginaw, Michigan
  - Troy, Michigan
  - Warren, Michigan
  - Golden Valley, Minnesota
  - Minneapolis, Minnesota
  - Saint Paul, Minnesota
  - Biloxi, Mississippi
  - Chesterfield, Missouri
  - Joplin, Missouri
  - Kansas City, Missouri
  - Saint Charles, Missouri
  - St Louis, Missouri
  - Kalispell, Montana
  - Fremont, Nebraska
  - Grand Island, Nebraska
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Henderson, Nevada
  - Belvidere, New Jersey
  - Brick, New Jersey
  - Bridgewater, New Jersey
  - Browns Mills, New Jersey
  - Cherry Hill, New Jersey
  - Elizabeth, New Jersey
  - Haddon Heights, New Jersey
  - Hamilton, New Jersey
  - Mine Hill, New Jersey
  - Ocean City, New Jersey
  - Passaic, New Jersey
  - Ridgewood, New Jersey
  - Somerset, New Jersey
  - Toms River, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Brooklyn, New York
  - Buffalo, New York
  - Cortlandt Manor, New York
  - Hawthorne, New York
  - Jamaica, New York
  - Mineola, New York
  - New York, New York
  - North Massapequa, New York
  - Saratoga Springs, New York
  - Troy, New York
  - Cary, North Carolina
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Greensboro, North Carolina
  - Mooresville, North Carolina
  - Morehead City, North Carolina
  - Morganton, North Carolina
  - Oxford, North Carolina
  - Pinehurst, North Carolina
  - Statesville, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Oakes, North Dakota
  - Akron, Ohio
  - Canal Fulton, Ohio
  - Canton, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Cuyahoga Falls, Ohio
  - Dayton, Ohio
  - Fairfield, Ohio
  - Marion, Ohio
  - Middletown, Ohio
  - Pitsburg, Ohio
  - Springfield, Ohio
  - Thornville, Ohio
  - Toledo, Ohio
  - Willoughby Hills, Ohio
  - Bartlesville, Oklahoma
  - Oklahoma City, Oklahoma
  - Bend, Oregon
  - Corvallis, Oregon
  - Altoona, Pennsylvania
  - Beaver, Pennsylvania
  - Chester, Pennsylvania
  - Clymer, Pennsylvania
  - Danville, Pennsylvania
  - Doylestown, Pennsylvania
  - Ephrata, Pennsylvania
  - Feasterville, Pennsylvania
  - Fleetwood, Pennsylvania
  - Greenville, Pennsylvania
  - Johnstown, Pennsylvania
  - Lancaster, Pennsylvania
  - Lewistown, Pennsylvania
  - Newport, Pennsylvania
  - Norristown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Pottstown, Pennsylvania
  - Scranton, Pennsylvania
  - Sellersville, Pennsylvania
  - Somerset, Pennsylvania
  - State College, Pennsylvania
  - Uniontown, Pennsylvania
  - Wilkes-Barre, Pennsylvania
  - Wynnewood, Pennsylvania
  - Yardley, Pennsylvania
  - Providence, Rhode Island
  - Anderson, South Carolina
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Florence, South Carolina
  - Greenville, South Carolina
  - Greer, South Carolina
  - Mt. Pleasant, South Carolina
  - Spartanburg, South Carolina
  - Summerville, South Carolina
  - Taylors, South Carolina
  - Walterboro, South Carolina
  - Rapid City, South Dakota
  - Columbia, Tennessee
  - Jackson, Tennessee
  - Johnson City, Tennessee
  - Nashville, Tennessee
  - Oak Ridge, Tennessee
  - Arlington, Texas
  - Austin, Texas
  - Carrollton, Texas
  - Corsicana, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Georgetown, Texas
  - Grapevine, Texas
  - Houston, Texas
  - Lubbock, Texas
  - McAllen, Texas
  - Odessa, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Tomball, Texas
  - Wichita Falls, Texas
  - Provo, Utah
  - West Valley City, Utah
  - Danville, Virginia
  - Hopewell, Virginia
  - Newport News, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Springfield, Virginia
  - Suffolk, Virginia
  - Virginia Beach, Virginia
  - Winchester, Virginia
  - Bellevue, Washington
  - Kirkland, Washington
  - Renton, Washington
  - Seattle, Washington
  - Spokane, Washington
  - Tacoma, Washington
  - Clarksburg, West Virginia
  - Madison, Wisconsin
  - Manitowoc, Wisconsin
  - Menomonee Falls, Wisconsin
- Argentina (17):
  - Bahía Blanca
  - Buenos Aires
  - Corrientes
  - Córdoba
  - Formosa
  - Godoy Cruz
  - Mar del Plata
  - Mendoza
  - Paraguay
  - Provincia de Chaco
  - Provincia de Rio Negro
  - Provincia de Salta
  - San Luis
  - San Miguel de Tucumán
  - San Salvador de Jujuy
  - Santa Fe
  - Sante Fe
- Australia (13):
  - Broken Hill, New South Wales
  - East Gosford, New South Wales
  - Carina Heights, Queensland
  - Milton, Queensland
  - Adelaide, South Australia
  - Frankston, Victoria
  - Ashford
  - Camperdown
  - Elizabeth Vale
  - Joondalup
  - Melbourne
  - Parkville
  - Perth
- Belgium (16):
  - Antwerp
  - Arlon
  - Bruges
  - Brussels
  - Genk
  - Hasselt
  - Leuven
  - Liège
  - Mechelen
  - Merksem
  - Moerkerke
  - Montegnée
  - Mousron
  - Torhout
  - Veurne
  - Wetteren
- Brazil (21):
  - Belo Horizonte
  - Blumenau
  - Brasília
  - Campina Grande do Sul
  - Campinas
  - Caxias do Sul
  - Curitiba
  - Goiânia
  - Lajeados
  - Maceió
  - Marília
  - Passo Fundo
  - Porto Alegre
  - Recife
  - Ribeirão Preto
  - Rio de Janeiro
  - Salvador
  - Santo André
  - São José
  - São Paulo
  - Uberlândia
- Bulgaria (8):
  - Burgas
  - Dimitrovgrad
  - Haskovo
  - Pleven
  - Plovdiv
  - Rousse
  - Sofia
  - Varna
- Canada (43):
  - Calgary, Alberta
  - Campbell River, British Columbia
  - Chilliwack, British Columbia
  - Coquitlam, British Columbia
  - Kamloops, British Columbia
  - Kelowna, British Columbia
  - New Westminster, British Columbia
  - Penticton, British Columbia
  - Quesnel, British Columbia
  - Victoria, British Columbia
  - Saint John, New Brunswick
  - Bridgewater, Nova Scotia
  - Halifax, Nova Scotia
  - Liverpool, Nova Scotia
  - Ajax, Ontario
  - Beamsville, Ontario
  - Brampton, Ontario
  - Corunna, Ontario
  - Greater Sudbury, Ontario
  - Hamilton, Ontario
  - Kitchener, Ontario
  - Listowel, Ontario
  - London, Ontario
  - Oshawa, Ontario
  - Ottawa, Ontario
  - Richmond Hill, Ontario
  - Sarnia, Ontario
  - Scarborough Village, Ontario
  - Toronto, Ontario
  - Greenfield Park, Quebec
  - Longueuil, Quebec
  - Montreal, Quebec
  - Québec, Quebec
  - Saint Georges de Beauce, Quebec
  - Saint-Charles-Borromée, Quebec
  - Saint-Jérôme, Quebec
  - Saint-Lambert, Quebec
  - Terrebonne, Quebec
  - Trois-Rivières, Quebec
  - Westmount, Quebec
  - Saskatoon, Saskatchewan
  - Mount Pearl
  - St. John's
- Chile (10):
  - Iquique
  - La Serena
  - Osorno
  - Port Montt
  - Rancagua
  - Santiago
  - Talcahuano
  - Temuco
  - Victoria
  - Viña del Mar
- China (22):
  - Baotou
  - Beijing
  - Changchun
  - Changsha
  - Chendu
  - Chongqing
  - Guangxi
  - Guangzhou
  - Hainan Province
  - Hangzhou
  - Harbin
  - Jinzhou
  - Lanzhou
  - Liaoning Province
  - Nanchang
  - Shaanxi Province
  - Shanghai
  - Shenyang
  - Shijiazhuang
  - Tianjin
  - Wenzhou
  - Wuhan
- Colombia (9):
  - Antioquia
  - Armenia
  - Barranquilla
  - Bogotá
  - Bucaramanga
  - Cartagena
  - Envigado
  - Manizales
  - Medellín
- Croatia (11):
  - Dubrovnik
  - Karlovac
  - Koprivnica
  - Krapinski Toplice
  - Osijek
  - Rijeka
  - Slavonski Brod
  - Split
  - Varaždin
  - Zadar
  - Zagreb
- Czechia (28):
  - Benátky nad Jizerou
  - Benešov
  - Bílovec
  - Brno
  - Brno-Lesna
  - Chrudim
  - Český Krumlov
  - Havlickux Brod
  - Hradec Králové
  - Hranice
  - Jindřichův Hradec
  - Kolín
  - Kroměříž
  - Mariánské Lázně
  - Mladá Boleslav
  - Náchod
  - Ostrava
  - Ostrava-Trebovice
  - Pardubice
  - Pilsen
  - Prague
  - Příbram
  - Řevnice
  - Semily
  - Slaný
  - Teplice
  - Trutnov
  - Ústí nad Labem
- Denmark (8):
  - Aarhus N
  - Copenhagen
  - Esbjerg
  - Frederiksberg
  - Glostrup Municipality
  - Hellerup
  - Holbæk
  - Horsens
- Estonia (5):
  - Haabneeme, Harju
  - Puusepa, Tartu
  - Pärnu
  - Tallinn
  - Tartu
- Finland (6):
  - Jyväskylä
  - Kuopio
  - Lappeenranta
  - Oulu
  - Seinäjoki
  - Tampere
- France (16):
  - Abbeville
  - Amiens
  - Brest
  - Cambrai
  - Clamart
  - La Roche-sur-Yon
  - Lille
  - Lyon
  - Massy
  - Nantes
  - Paris
  - Pau
  - Pessac
  - Poitiers
  - Tours
  - Valenciennes
- Germany (46):
  - Altenburg
  - Aschaffenburg
  - Augsburg
  - Bad Nauheim
  - Berlin
  - Bochum
  - Cloppenburg
  - Cologne
  - Dortmund
  - Dresden
  - Essen
  - Frankfurt
  - Giengen an der Brenz
  - Görlitz
  - Großheirath
  - Hamburg
  - Heidelberg
  - Heilbronn
  - Homburg
  - Ingelheim
  - Kallstadt
  - Kassel
  - Kiel-Kronshagen
  - Leipzig
  - Ludwigshafen
  - Lübeck
  - Magdeburg
  - Mainz
  - Mannheim
  - Markkleeberg
  - München
  - Nienburg
  - Northeinm
  - Offenbach-beiber
  - Potsdam
  - Rüdersdorf
  - Siegen
  - Stuhr
  - Ulm
  - Unterschneidheim
  - Wardenburg
  - Wermsdorf
  - Weyhe
  - Witten
  - Woerishofen
  - Wuppertal
- Greece (7):
  - Athens
  - Larissa
  - Rhodes
  - Rio-Patras
  - Thessaloniki
  - Trikala
  - Voula
- Guatemala (7):
  - Ciudad
  - Clinica
  - Edificio Multimedica
  - Nivel
  - Oficina
  - Quetzaltenango
  - Zacapa
- Hungary (18):
  - Ajka
  - Baja
  - Békéscsaba
  - Budapest
  - Debrecen
  - Hódmezővásárhely
  - Kecskemét
  - Keeskemet
  - Kistarcsa
  - Komárom
  - Makó
  - Nagykanizsa
  - Nyíregyháza
  - Pécs
  - Sopron
  - Szekszárd
  - Szombathely
  - Zalaegerszeg
- India (37):
  - Hyderabad, Andhra Pradesh
  - Vijayawada, Andhra Pradesh
  - Angamaly, Kerala
  - Kochi, Kerala
  - Thrissur, Kerala
  - Ahmedabad
  - Anddhra Pradesh
  - Andhra Pradesh
  - Aurangabad
  - Bangalore
  - Bikaner
  - Chennai
  - Coimbatore
  - Delhi
  - Gujrāt
  - Indore
  - Jaipur
  - Karnataka
  - Kerala
  - Kolkata
  - Ludhiana
  - Madhya Pradesh
  - Maharashtra
  - Mangalore
  - Mumbai
  - Nagpur
  - Nashik
  - New Delhi
  - Pune
  - Punjab
  - Pūni
  - Rajasthan
  - Ramnagar
  - Shimoga
  - Surat
  - Trivandrum
  - Vadodara
- Israel (18):
  - Afula
  - Beersheba
  - Dimona
  - Giv‘atayim
  - Hadera
  - Haifa
  - Holon
  - Jerusalem
  - Kfar Saba
  - Nahariya
  - Nazareth
  - Petah Tikva
  - Poria – Neve Oved
  - Raanana
  - Rehovot
  - Tel Aviv
  - Tel Litwinsky
  - Ẕerifin
- Italy (26):
  - Bologna
  - Brescia
  - Cantania
  - Casarano
  - Caserta
  - Chieti
  - Cremona
  - Genova
  - Grosseto
  - Legnano
  - Manerbio
  - Milan
  - Monserrato
  - Napoli
  - Novara
  - Ostia Antica
  - Pavia
  - Pisa
  - Pozzuoli
  - Roma
  - Santa Maria Capua Vetere
  - Sassari
  - Seriate
  - Siena
  - Trieste
  - Venezia Mestre
- Japan (39):
  - Kyoto, Kyoto
  - Lida-shi, Nagano
  - Ueda-shi, Nagano
  - Minato-ku, Tokyo
  - Aichi
  - Aomori
  - Chiaki
  - Chiba
  - Ehime
  - Fukuoka
  - Fukushima
  - Gifu
  - Gunma
  - Hiroshima
  - Hokkai-do
  - Hokkaido
  - Hyōgo
  - Ibaraki
  - Isesaki-shi
  - Ishikawa
  - Kagawa
  - Kanagawa
  - Kumamoto
  - Kyoda
  - Mie
  - Miyagi
  - Nagaoka-shi
  - Nagasaki
  - Niigata
  - Numakunai
  - Okayama
  - Osaka
  - Saitama
  - Shimane
  - Shizuoka
  - Tokushima
  - Tokyo
  - Yamaguchi
  - Yokohama
- Mexico (9):
  - Guadalajara, Jalisco
  - Xalapa, Veracruz
  - Aguascalientes
  - Chihuahua City
  - Distrito Federal
  - Durango
  - Monterrey
  - San Luis Potosí City
  - Yucatán
- Netherlands (11):
  - Almere Stad
  - Amstelveen
  - Amsterdam
  - Dordrecht
  - Eindhoven
  - Ewijk
  - Leiderdorp
  - Maastricht
  - Rotterdam
  - Venlo
  - Wildervlank
- New Zealand (7):
  - Lower Hutt, Wellington Region
  - Auckland
  - Christchurch
  - Dunedin
  - Hamilton
  - Nelson
  - Tauranga
- Norway (5):
  - Bodø
  - Harstad
  - Haugesund
  - Oslo
  - Rud
- Peru (3):
  - Arequipa
  - Callao
  - Lima
- Philippines (5):
  - Cebu
  - Cebu City
  - Davao City
  - Pasig
  - Quezon City
- Poland (31):
  - Ostrów, Mazowiecka
  - Bydgoszcz
  - Chojnice
  - Elblag
  - Ełk
  - Gdansk
  - Inowrocław
  - Jarosław
  - Katowice
  - Komenskiego
  - Kołobrzeg
  - Krakow
  - Kutno
  - Libiąż
  - Lodz
  - Lubartów
  - Lublin
  - Pomorskie
  - Puławy
  - Płock
  - Ruda Śląska
  - Rzeszów
  - Skierniewice
  - Sopot
  - Sucharskiego
  - Szczecin
  - Tarnów
  - Torun
  - Warsaw
  - Warzawa
  - Wroclaw
- Portugal (9):
  - Amadora
  - Aveiro
  - Braga
  - Coimbra
  - Leiria
  - Lisbon
  - Ponta Delgada
  - Setúbal
  - Viseu
- Romania (15):
  - Bacau
  - Brasov
  - Brăila
  - Buccuresti
  - Bucharest
  - Buzău
  - Covasna
  - Dambovita
  - Iași
  - Judetul Maramures
  - Judetul Mures
  - Judetul Suceava
  - Judetul Vrancea
  - Oradea
  - Timișoara
- Russia (19):
  - Barnaul
  - Chelyabinsk
  - Kemerovo
  - Krasnoyarsk
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - Omsk
  - Orenburg
  - Perm
  - Ryazan
  - Saint Petersburg
  - Saratov
  - Smolensk
  - Tula
  - Tyumen
  - Volgograd
  - Voronezh
  - Yaroslavl
- Serbia (6):
  - Belgrade
  - Kamenitz
  - Niš
  - Niška Banja
  - Zemun
  - Zmaj Jovina
- Slovakia (11):
  - Bardejov
  - Bratislava
  - Dolný Kubín
  - Galanta
  - Košice
  - Levice
  - Lučenec
  - Nitra
  - Nové Zámky
  - Prešov
  - Rimavská Sobota
- South Africa (13):
  - Alberton
  - Benoni
  - Bloemfontein
  - Cape Town
  - Diepkloof
  - Durban
  - Lyttelton
  - Parktown West
  - Port Elizabeth
  - Potchefstroom
  - Pretoria
  - Somerset West
  - Worcester
- South Korea (9):
  - Busan
  - Daegu
  - Daejeon
  - Gangwon-do
  - Gwangju
  - Gyeonggi-do
  - Incheon
  - Pusan
  - Seoul
- Spain (16):
  - A Coruña
  - Alcoy
  - Almería
  - Barcelona
  - Bilbao
  - De La Castellana
  - Donostia / San Sebastian
  - Figueras
  - Jaén
  - Lleida
  - Madrid
  - Murcia
  - Santiago de Compostela
  - Seville
  - Vigo
  - Vitoria-Gasteiz
- Sweden (17):
  - Alingsås
  - Enköping
  - Gothenburg
  - Halmstad
  - Karlshamn
  - Köping
  - Lindesberg
  - Luleå
  - Lund
  - Malmo
  - Mora
  - Mölndal
  - Örebro
  - Skene
  - Umeå
  - Uppsala
  - Varberg
- Switzerland (2):
  - Lausanne
  - Lugano
- Taiwan (7):
  - Changhua
  - Hualien City
  - Kaohsiung City
  - Taichung
  - Taipei
  - Taoyuan
  - Yongkang District
- Thailand (7):
  - Bangkok
  - Chang Mai
  - Khon Kaen
  - Nakhon Ratchasima
  - Pathum Thani
  - Sai Mai
  - Songkhla
- Turkey (Türkiye) (11):
  - Adana
  - Ankara
  - Antalya
  - Aydin
  - Erzurum
  - Eskişehir
  - Isparta
  - Istanbul
  - Izmir
  - Konya
  - Sivas
- Ukraine (18):
  - Cherkasy
  - Chernihiv
  - Dnipropetrovsk
  - Donetsk
  - Ivano-Frankivsh
  - Ivano-Frankivsk
  - Kharkiv
  - Kherson
  - Kyiv
  - Luhansk
  - Lutsk
  - Lviv
  - Mykolayiv
  - Odesa
  - Poltava
  - Uzhhorod
  - Vinnytsia
  - Zaporizhzhya
- United Kingdom (31):
  - Birmingham
  - Blackpool
  - Bournemouth
  - Bradford
  - Cambridge
  - Chesterfield
  - Coventry
  - Devon
  - Dundee
  - East Horsley
  - East Sussex
  - Edinburgh
  - Essex
  - Glasgow
  - Harrow
  - Leicester
  - Liverpool
  - London
  - Middlesbrough
  - Orpington
  - Peterborough
  - Portadown
  - Sheffield
  - Stirling
  - Stockport
  - Surrey
  - Sutton Coldfield
  - Swindon
  - Warwickshire
  - Wolverhampton
  - York

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Semco RS, Bergmark RW, Murphy SA, Cange AL, Unverdorben M, Chen CZL, Ruff CT, Antman EM, Giugliano RP, Bergmark BA. Epistaxis Versus Nonepistaxis Bleeding in Anticoagulated Patients With Atrial Fibrillation: Results From the ENGAGE AF-TIMI 48 Trial. J Am Heart Assoc. 2025 Jan 21;14(2):e031434. doi: 10.1161/JAHA.123.031434. Epub 2025 Jan 10. PMID 39791401
- [Derived] Zimerman A, Braunwald E, Steffel J, Van Mieghem NM, Palazzolo MG, Murphy SA, Chen CZL, Unverdorben M, Ruff CT, Antman EM, Giugliano RP. Dose Reduction of Edoxaban in Patients 80 Years and Older With Atrial Fibrillation: Post Hoc Analysis of the ENGAGE AF-TIMI 48 Randomized Clinical Trial. JAMA Cardiol. 2024 Sep 1;9(9):817-825. doi: 10.1001/jamacardio.2024.1793. PMID 38985461
- [Derived] Bergmark BA, Park JG, Hamershock RA, Melloni GEM, De Caterina R, Antman EM, Ruff CT, Rutman H, Mercuri MF, Lanz HJ, Braunwald E, Giugliano RP. Application of the Win Ratio Method in the ENGAGE AF-TIMI 48 Trial Comparing Edoxaban With Warfarin in Patients With Atrial Fibrillation. Circ Cardiovasc Qual Outcomes. 2024 Jul;17(7):e010561. doi: 10.1161/CIRCOUTCOMES.123.010561. Epub 2024 Jun 3. PMID 38828563
- [Derived] Inciardi RM, Giugliano RP, Park JG, Nordio F, Ruff CT, Chen C, Lanz HJ, Antman EM, Braunwald E, Solomon SD. Risks of Heart Failure, Stroke, and Bleeding in Atrial Fibrillation According to Heart Failure Phenotypes. JACC Clin Electrophysiol. 2023 Apr;9(4):569-580. doi: 10.1016/j.jacep.2022.11.032. Epub 2023 Feb 22. PMID 37100536
- [Derived] Oyama K, Giugliano RP, Ruff CT, Berg DD, Jarolim P, Tang M, Park JG, Lanz HJ, Antman EM, Braunwald E, Morrow DA. Serial assessment of biomarkers and heart failure outcomes in patients with atrial fibrillation. Eur J Heart Fail. 2023 Jun;25(6):832-841. doi: 10.1002/ejhf.2844. Epub 2023 Apr 18. PMID 36987929
- [Derived] Bonaca MP, Antman EM, Cunningham JW, Wiviott SD, Murphy SA, Halperin JL, Weitz JI, Grosso MA, Lanz HJ, Braunwald E, Giugliano RP, Ruff CT. Ischaemic and bleeding risk in atrial fibrillation with and without peripheral artery disease and efficacy and safety of full- and half-dose edoxaban vs. warfarin: insights from ENGAGE AF-TIMI 48. Eur Heart J Cardiovasc Pharmacother. 2022 Sep 29;8(7):695-706. doi: 10.1093/ehjcvp/pvab089. PMID 34962979
- [Derived] Oyama K, Giugliano RP, Berg DD, Ruff CT, Jarolim P, Tang M, Murphy SA, Lanz HJ, Grosso MA, Antman EM, Braunwald E, Morrow DA. Serial assessment of biomarkers and the risk of stroke or systemic embolism and bleeding in patients with atrial fibrillation in the ENGAGE AF-TIMI 48 trial. Eur Heart J. 2021 May 1;42(17):1698-1706. doi: 10.1093/eurheartj/ehab141. PMID 33760027
- [Derived] Steffel J, Ruff CT, Yin O, Braunwald E, Park JG, Murphy SA, Connolly S, Antman EM, Giugliano RP. Randomized, Double-Blind Comparison of Half-Dose Versus Full-Dose Edoxaban in 14,014 Patients With Atrial Fibrillation. J Am Coll Cardiol. 2021 Mar 9;77(9):1197-1207. doi: 10.1016/j.jacc.2020.12.053. PMID 33663737
- [Derived] Wilkinson C, Wu J, Searle SD, Todd O, Hall M, Kunadian V, Clegg A, Rockwood K, Gale CP. Clinical outcomes in patients with atrial fibrillation and frailty: insights from the ENGAGE AF-TIMI 48 trial. BMC Med. 2020 Dec 24;18(1):401. doi: 10.1186/s12916-020-01870-w. PMID 33357217
- [Derived] Vilain K, Li H, Kwong WJ, Antman EM, Ruff CT, Braunwald E, Cohen DJ, Giugliano RP, Magnuson EA; ENGAGE AF-TIMI 48 Trial Investigators. Cardiovascular- and Bleeding-Related Hospitalization Rates With Edoxaban Versus Warfarin in Patients With Atrial Fibrillation Based on Results of the ENGAGE AF-TIMI 48 Trial. Circ Cardiovasc Qual Outcomes. 2020 Nov;13(11):e006511. doi: 10.1161/CIRCOUTCOMES.120.006511. Epub 2020 Nov 5. PMID 33148013
- [Derived] Inciardi RM, Giugliano RP, Claggett B, Gupta DK, Chandra A, Ruff CT, Antman EM, Mercuri MF, Grosso MA, Braunwald E, Solomon SD; ENGAGE AF-TIMI 48 Investigators. Left atrial structure and function and the risk of death or heart failure in atrial fibrillation. Eur J Heart Fail. 2019 Dec;21(12):1571-1579. doi: 10.1002/ejhf.1606. Epub 2019 Nov 27. PMID 31777160
- [Derived] Bergmark BA, Kamphuisen PW, Wiviott SD, Ruff CT, Antman EM, Nordio F, Kuder JF, Mercuri MF, Lanz HJ, Braunwald E, Giugliano RP. Comparison of Events Across Bleeding Scales in the ENGAGE AF-TIMI 48 Trial. Circulation. 2019 Nov 26;140(22):1792-1801. doi: 10.1161/CIRCULATIONAHA.119.041346. Epub 2019 Oct 10. PMID 31597460
- [Derived] Berg DD, Ruff CT, Jarolim P, Giugliano RP, Nordio F, Lanz HJ, Mercuri MF, Antman EM, Braunwald E, Morrow DA. Performance of the ABC Scores for Assessing the Risk of Stroke or Systemic Embolism and Bleeding in Patients With Atrial Fibrillation in ENGAGE AF-TIMI 48. Circulation. 2019 Feb 5;139(6):760-771. doi: 10.1161/CIRCULATIONAHA.118.038312. PMID 30586727
- [Derived] Corbalan R, Nicolau JC, Lopez-Sendon J, Garcia-Castillo A, Botero R, Sotomora G, Horna M, Ruff CT, Hamershock RA, Grip LT, Antman EM, Braunwald E, Giugliano RP. Edoxaban Versus Warfarin in Latin American Patients With Atrial Fibrillation: The ENGAGE AF-TIMI 48 Trial. J Am Coll Cardiol. 2018 Sep 25;72(13):1466-1475. doi: 10.1016/j.jacc.2018.07.037. PMID 30236308
- [Derived] Yin OQP, Antman EM, Braunwald E, Mercuri MF, Miller R, Morrow D, Ruff CT, Truitt K, Weitz JI, Giugliano RP. Linking Endogenous Factor Xa Activity, a Biologically Relevant Pharmacodynamic Marker, to Edoxaban Plasma Concentrations and Clinical Outcomes in the ENGAGE AF-TIMI 48 Trial. Circulation. 2018 Oct 30;138(18):1963-1973. doi: 10.1161/CIRCULATIONAHA.118.033933. PMID 29967197
- [Derived] Aisenberg J, Chatterjee-Murphy P, Friedman Flack K, Weitz JI, Ruff CT, Nordio F, Mercuri MF, Choi Y, Antman EM, Braunwald E, Giugliano RP. Gastrointestinal Bleeding With Edoxaban Versus Warfarin: Results From the ENGAGE AF-TIMI 48 Trial (Effective Anticoagulation With Factor Xa Next Generation in Atrial Fibrillation-Thrombolysis In Myocardial Infarction). Circ Cardiovasc Qual Outcomes. 2018 May;11(5):e003998. doi: 10.1161/CIRCOUTCOMES.117.003998. PMID 29748353
- [Derived] Wang K, Li H, Kwong WJ, Antman EM, Ruff CT, Giugliano RP, Cohen DJ, Magnuson EA; ENGAGE AF-TIMI 48 Trial Investigators. Impact of Spontaneous Extracranial Bleeding Events on Health State Utility in Patients with Atrial Fibrillation: Results from the ENGAGE AF-TIMI 48 Trial. J Am Heart Assoc. 2017 Aug 11;6(8):e006703. doi: 10.1161/JAHA.117.006703. PMID 28862934
- [Derived] Eisen A, Ruff CT, Braunwald E, Hamershock RA, Lewis BS, Hassager C, Chao TF, Le Heuzey JY, Mercuri M, Rutman H, Antman EM, Giugliano RP. Digoxin Use and Subsequent Clinical Outcomes in Patients With Atrial Fibrillation With or Without Heart Failure in the ENGAGE AF-TIMI 48 Trial. J Am Heart Assoc. 2017 Jun 30;6(7):e006035. doi: 10.1161/JAHA.117.006035. PMID 28666993
- [Derived] De Caterina R, Renda G, Carnicelli AP, Nordio F, Trevisan M, Mercuri MF, Ruff CT, Antman EM, Braunwald E, Giugliano RP. Valvular Heart Disease Patients on Edoxaban or Warfarin in the ENGAGE AF-TIMI 48 Trial. J Am Coll Cardiol. 2017 Mar 21;69(11):1372-1382. doi: 10.1016/j.jacc.2016.12.031. PMID 28302288
- [Derived] Link MS, Giugliano RP, Ruff CT, Scirica BM, Huikuri H, Oto A, Crompton AE, Murphy SA, Lanz H, Mercuri MF, Antman EM, Braunwald E; ENGAGE AF-TIMI 48 Investigators. Stroke and Mortality Risk in Patients With Various Patterns of Atrial Fibrillation: Results From the ENGAGE AF-TIMI 48 Trial (Effective Anticoagulation With Factor Xa Next Generation in Atrial Fibrillation-Thrombolysis in Myocardial Infarction 48). Circ Arrhythm Electrophysiol. 2017 Jan;10(1):e004267. doi: 10.1161/CIRCEP.116.004267. PMID 28077507
- [Derived] Ruff CT, Giugliano RP, Braunwald E, Murphy SA, Brown K, Jarolim P, Mercuri M, Antman EM, Morrow DA. Cardiovascular Biomarker Score and Clinical Outcomes in Patients With Atrial Fibrillation: A Subanalysis of the ENGAGE AF-TIMI 48 Randomized Clinical Trial. JAMA Cardiol. 2016 Dec 1;1(9):999-1006. doi: 10.1001/jamacardio.2016.3311. PMID 27706467
- [Derived] Steffel J, Giugliano RP, Braunwald E, Murphy SA, Mercuri M, Choi Y, Aylward P, White H, Zamorano JL, Antman EM, Ruff CT. Edoxaban Versus Warfarin in Atrial Fibrillation Patients at Risk of Falling: ENGAGE AF-TIMI 48 Analysis. J Am Coll Cardiol. 2016 Sep 13;68(11):1169-1178. doi: 10.1016/j.jacc.2016.06.034. PMID 27609678
- [Derived] Eisen A, Ruff CT, Braunwald E, Nordio F, Corbalan R, Dalby A, Dorobantu M, Mercuri M, Lanz H, Rutman H, Wiviott SD, Antman EM, Giugliano RP. Sudden Cardiac Death in Patients With Atrial Fibrillation: Insights From the ENGAGE AF-TIMI 48 Trial. J Am Heart Assoc. 2016 Jul 8;5(7):e003735. doi: 10.1161/JAHA.116.003735. PMID 27402235
- [Derived] Rost NS, Giugliano RP, Ruff CT, Murphy SA, Crompton AE, Norden AD, Silverman S, Singhal AB, Nicolau JC, SomaRaju B, Mercuri MF, Antman EM, Braunwald E; ENGAGE AF-TIMI 48 Investigators. Outcomes With Edoxaban Versus Warfarin in Patients With Previous Cerebrovascular Events: Findings From ENGAGE AF-TIMI 48 (Effective Anticoagulation With Factor Xa Next Generation in Atrial Fibrillation-Thrombolysis in Myocardial Infarction 48). Stroke. 2016 Aug;47(8):2075-82. doi: 10.1161/STROKEAHA.116.013540. Epub 2016 Jul 7. PMID 27387994
- [Derived] Bohula EA, Giugliano RP, Ruff CT, Kuder JF, Murphy SA, Antman EM, Braunwald E. Impact of Renal Function on Outcomes With Edoxaban in the ENGAGE AF-TIMI 48 Trial. Circulation. 2016 Jul 5;134(1):24-36. doi: 10.1161/CIRCULATIONAHA.116.022361. PMID 27358434
- [Derived] Kato ET, Giugliano RP, Ruff CT, Koretsune Y, Yamashita T, Kiss RG, Nordio F, Murphy SA, Kimura T, Jin J, Lanz H, Mercuri M, Braunwald E, Antman EM. Efficacy and Safety of Edoxaban in Elderly Patients With Atrial Fibrillation in the ENGAGE AF-TIMI 48 Trial. J Am Heart Assoc. 2016 May 20;5(5):e003432. doi: 10.1161/JAHA.116.003432. PMID 27207971
- [Derived] Xu H, Ruff CT, Giugliano RP, Murphy SA, Nordio F, Patel I, Shi M, Mercuri M, Antman EM, Braunwald E. Concomitant Use of Single Antiplatelet Therapy With Edoxaban or Warfarin in Patients With Atrial Fibrillation: Analysis From the ENGAGE AF-TIMI48 Trial. J Am Heart Assoc. 2016 Feb 23;5(2):e002587. doi: 10.1161/JAHA.115.002587. PMID 26908401
- [Derived] Ruff CT, Giugliano RP, Braunwald E, Morrow DA, Murphy SA, Kuder JF, Deenadayalu N, Jarolim P, Betcher J, Shi M, Brown K, Patel I, Mercuri M, Antman EM. Association between edoxaban dose, concentration, anti-Factor Xa activity, and outcomes: an analysis of data from the randomised, double-blind ENGAGE AF-TIMI 48 trial. Lancet. 2015 Jun 6;385(9984):2288-95. doi: 10.1016/S0140-6736(14)61943-7. Epub 2015 Mar 11. PMID 25769361
- [Derived] Mega JL, Walker JR, Ruff CT, Vandell AG, Nordio F, Deenadayalu N, Murphy SA, Lee J, Mercuri MF, Giugliano RP, Antman EM, Braunwald E, Sabatine MS. Genetics and the clinical response to warfarin and edoxaban: findings from the randomised, double-blind ENGAGE AF-TIMI 48 trial. Lancet. 2015 Jun 6;385(9984):2280-7. doi: 10.1016/S0140-6736(14)61994-2. Epub 2015 Mar 11. PMID 25769357
- [Derived] Ruff CT, Giugliano RP, Braunwald E, Mercuri M, Curt V, Betcher J, Grip L, Cange AL, Crompton AE, Murphy SA, Deenadayalu N, Antman EM. Transition of patients from blinded study drug to open-label anticoagulation: the ENGAGE AF-TIMI 48 trial. J Am Coll Cardiol. 2014 Aug 12;64(6):576-84. doi: 10.1016/j.jacc.2014.05.028. PMID 25104527
- [Derived] Giugliano RP, Ruff CT, Rost NS, Silverman S, Wiviott SD, Lowe C, Deenadayalu N, Murphy SA, Grip LT, Betcher JM, Duggal A, Dave J, Shi M, Mercuri M, Antman EM, Braunwald E; ENGAGE AF-TIMI 48 Investigators. Cerebrovascular events in 21 105 patients with atrial fibrillation randomized to edoxaban versus warfarin: Effective Anticoagulation with Factor Xa Next Generation in Atrial Fibrillation-Thrombolysis in Myocardial Infarction 48. Stroke. 2014 Aug;45(8):2372-8. doi: 10.1161/STROKEAHA.114.006025. Epub 2014 Jun 19. PMID 24947287
- [Derived] Gupta DK, Shah AM, Giugliano RP, Ruff CT, Antman EM, Grip LT, Deenadayalu N, Hoffman E, Patel I, Shi M, Mercuri M, Mitrovic V, Braunwald E, Solomon SD; Effective aNticoaGulation with factor xA next GEneration in AF-Thrombolysis In Myocardial Infarction 48 Echocardiographic Study Investigators. Left atrial structure and function in atrial fibrillation: ENGAGE AF-TIMI 48. Eur Heart J. 2014 Jun 7;35(22):1457-65. doi: 10.1093/eurheartj/eht500. Epub 2013 Dec 2. PMID 24302269
- [Derived] Giugliano RP, Ruff CT, Braunwald E, Murphy SA, Wiviott SD, Halperin JL, Waldo AL, Ezekowitz MD, Weitz JI, Spinar J, Ruzyllo W, Ruda M, Koretsune Y, Betcher J, Shi M, Grip LT, Patel SP, Patel I, Hanyok JJ, Mercuri M, Antman EM; ENGAGE AF-TIMI 48 Investigators. Edoxaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2013 Nov 28;369(22):2093-104. doi: 10.1056/NEJMoa1310907. Epub 2013 Nov 19. PMID 24251359
- [Derived] Salazar DE, Mendell J, Kastrissios H, Green M, Carrothers TJ, Song S, Patel I, Bocanegra TS, Antman EM, Giugliano RP, Kunitada S, Dornseif B, Shi M, Tachibana M, Zhou S, Rohatagi S. Modelling and simulation of edoxaban exposure and response relationships in patients with atrial fibrillation. Thromb Haemost. 2012 May;107(5):925-36. doi: 10.1160/TH11-08-0566. Epub 2012 Mar 8. PMID 22398655
- [Derived] Ruff CT, Giugliano RP, Antman EM, Crugnale SE, Bocanegra T, Mercuri M, Hanyok J, Patel I, Shi M, Salazar D, McCabe CH, Braunwald E. Evaluation of the novel factor Xa inhibitor edoxaban compared with warfarin in patients with atrial fibrillation: design and rationale for the Effective aNticoaGulation with factor xA next GEneration in Atrial Fibrillation-Thrombolysis In Myocardial Infarction study 48 (ENGAGE AF-TIMI 48). Am Heart J. 2010 Oct;160(4):635-41. doi: 10.1016/j.ahj.2010.06.042. PMID 20934556

RESULTS

PARTICIPANT FLOW:
Groups:
- High Dose Edoxaban/Placebo Warfarin: Edoxaban tablets plus warfarin placebo tablets
  60mg Edoxaban tablets (high dose regimen): Edoxaban tablets plus warfarin placebo tablets each taken once daily for 24 months
  placebo warfarin: placebo warfarin
- Low Dose Edoxaban/Placebo Warfarin: Edoxaban tablets plus warfarin placebo tablets
  30mg Edoxaban tablets (low dose regimen): Edoxaban tablets plus warfarin placebo tablets each taken once daily for 24 months
  placebo warfarin: placebo warfarin
Period: Overall Study
Arm/Group | Warfarin/Placebo Edoxaban | High Dose Edoxaban/Placebo Warfarin | Low Dose Edoxaban/Placebo Warfarin
Started | 7036 | 7035 | 7034
Safety Analysis Set (Received Drug) | 7012 | 7012 | 7002
mITT Analysis Set (Received Drug) | 7012 | 7012 | 7002
Per Protocol Analysis Set | 6993 | 6995 | 6982
Completed | 6157 | 6228 | 6250
Not Completed | 879 | 807 | 784
Not completed — never received study drug | 24 | 23 | 32
Not completed — Protocol Violation | 19 | 17 | 20
Not completed — Death | 789 | 730 | 706
Not completed — Withdrawal by Subject | 47 | 37 | 25
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Warfarin/Placebo Edoxaban | High Dose Edoxaban/Placebo Warfarin | Low Dose Edoxaban/Placebo Warfarin | Total
Number analyzed (Participants) | 7012 | 7012 | 7002 | 21026
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1869 | 1830 | 1784 | 5483
  >=65 years | 5143 | 5182 | 5218 | 15543
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.5 (9.44) | 70.6 (9.51) | 70.6 (9.31) | 70.6 (9.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2629 | 2659 | 2718 | 8006
  Male | 4383 | 4353 | 4284 | 13020
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 963 | 956 | 975 | 2894
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 88 | 96 | 94 | 278
  White | 5679 | 5679 | 5650 | 17008
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 282 | 281 | 283 | 846
Region of Enrollment [Number; unit: participants]
  Portugal | 46 | 71 | 61 | 178
  United States | 1297 | 1288 | 1308 | 3893
  Serbia | 95 | 107 | 74 | 276
  Philippines | 43 | 36 | 45 | 124
  Estonia | 76 | 55 | 60 | 191
  Taiwan | 77 | 72 | 85 | 234
  Slovakia | 143 | 133 | 129 | 405
  Greece | 14 | 27 | 9 | 50
  Spain | 44 | 65 | 54 | 163
  Thailand | 40 | 40 | 33 | 113
  Ukraine | 360 | 386 | 402 | 1148
  Israel | 104 | 88 | 88 | 280
  Chile | 74 | 91 | 88 | 253
  Russian Federation | 375 | 406 | 369 | 1150
  Colombia | 51 | 42 | 48 | 141
  Switzerland | 0 | 1 | 4 | 5
  Italy | 60 | 55 | 54 | 169
  India | 232 | 220 | 234 | 686
  France | 40 | 38 | 32 | 110
  Peru | 64 | 46 | 60 | 170
  Denmark | 68 | 80 | 70 | 218
  Australia | 30 | 40 | 32 | 102
  South Africa | 97 | 92 | 90 | 279
  Netherlands | 64 | 49 | 40 | 153
  China | 163 | 150 | 152 | 465
  Korea, Republic of | 64 | 84 | 78 | 226
  Finland | 9 | 18 | 15 | 42
  Guatemala | 48 | 48 | 39 | 135
  Turkey | 40 | 39 | 31 | 110
  United Kingdom | 132 | 121 | 145 | 398
  Hungary | 151 | 143 | 167 | 461
  Czech Republic | 410 | 369 | 386 | 1165
  Mexico | 60 | 70 | 60 | 190
  Canada | 259 | 271 | 242 | 772
  Argentina | 352 | 345 | 362 | 1059
  Brazil | 236 | 242 | 225 | 703
  Belgium | 41 | 44 | 64 | 149
  Poland | 395 | 424 | 454 | 1273
  Croatia | 53 | 33 | 39 | 125
  Romania | 141 | 144 | 124 | 409
  Bulgaria | 179 | 174 | 165 | 518
  Norway | 11 | 8 | 15 | 34
  Germany | 308 | 293 | 307 | 908
  Japan | 337 | 336 | 337 | 1010
  New Zealand | 40 | 50 | 40 | 130
  Sweden | 89 | 78 | 86 | 253

OUTCOME MEASURES:

1. Primary Outcome: Compare Edoxaban to Warfarin for Composite of Stroke and Systemic Embolic Events (SEE).
Description: The composite of stroke and Systemic Embolic Events (SEE) during the on treatment period in the mITT analysis population with a non-inferiority analysis.
Time Frame: on-treatment period 2.5 years of median study drug exposure and 2.8 year of median follow-up
Population: mITT (modified Intent To Treat) Analysis set; which included randomized subjects who received 1 or more dose of study drug. The time period included the subject was taking study drug and up to 3 days after their last dose (On-Treatment ).
Measure: Number; unit: number of participants with event
Arm/Group | Low Dose Edoxaban/Placebo Warfarin | High Dose Edoxaban/Placebo Warfarin | Warfarin/Placebo Edoxaban
Number analyzed (Participants) | 7002 | 7012 | 7012
number of participants with event | 253 | 182 | 232
Statistical Analysis 1: Comparison: High Dose Edoxaban/Placebo Warfarin vs Warfarin/Placebo Edoxaban; The primary efficacy endpoint, time to the first occurrence of stroke/SEE, was first compared concurrently between each of the 2 edoxaban groups and warfarin group using the mITT Analysis Set in the on-treatment period for non-inferiority. In order to control the study-wise type-I error rate of two-sided α=0.05 for non-inferiority, each of these 2 comparisons were performed at the statistical significance level of two-sided α=0.025, respectively; Test type: Non-Inferiority or Equivalence — The non-inferiority analysis included the mITT and PP analysis sets for both the on treatment and overall study period, although mITT on-treatment was considered primary; p < .0001, Cox proportional hazards model — Two stratification factor covariates: 1) CHADS2 score 2) dose-adjustment factor. If upper limit of CI of HR was below 1.38, then non-inferiority to warfarin was established for group; Hazard Ratio (HR) = 0.79, 97.5% CI 2-sided [.632 to .985]
Statistical Analysis 2: Comparison: Low Dose Edoxaban/Placebo Warfarin vs Warfarin/Placebo Edoxaban; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = .0055, Cox proportional hazards model — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.07, 97.5% CI 2-sided [.874 to 1.314]

2. Primary Outcome: Compare Edoxaban to Warfarin for Composite of Stroke and Systemic Embolic Events (SEE).
Description: The composite of stroke and Systemic Embolic Events (SEE) during the overall study period in the mITT analysis population.
Time Frame: overall study period 2.5 years of median study drug exposure and 2.8 year of median follow-up
Population: mITT (modified Intent To Treat) Analysis set; which included randomized subjects who received 1 or more dose of study drug. The time frame included overall study period (first dose to end of study).
Measure: Number; unit: Number of participants with event
Arm/Group | Low Dose Edoxaban/Placebo Warfarin | High Dose Edoxaban/Placebo Warfarin | Warfarin/Placebo Edoxaban
Number analyzed (Participants) | 7002 | 7012 | 7012
Number of participants with event | 382 | 292 | 336
Statistical Analysis 1: Comparison: High Dose Edoxaban/Placebo Warfarin vs Warfarin/Placebo Edoxaban; Non-inferiority or equivalence analysis; Non-inferiority analysis. The non-inferiority analysis included the mITT and PP analysis sets for both the on treatment and overall study period, although mITT on-treatment was considered primary; Test type: Non-Inferiority or Equivalence — If the upper limit of this CI of the hazard ratio was below 1.38, then non-inferiority to warfarin was considered established for the edoxaban treatment group; p < .0001, Cox proportional hazards model; Hazard Ratio (HR) = .86, 97.5% CI 2-sided [.719 to 1.029]
Statistical Analysis 2: Comparison: Low Dose Edoxaban/Placebo Warfarin vs Warfarin/Placebo Edoxaban; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = .0074, Cox proportional hazards model; Hazard Ratio (HR) = 1.13, 97.5% CI 2-sided [.955 to 1.336]

3. Primary Outcome: Compare Edoxaban to Warfarin for Composite of Stroke and Systemic Embolic Events (SEE).
Description: The composite of stroke and Systemic Embolic Events (SEE) during the on treatment period in the PP (per protocol) analysis set population.
Time Frame: on-treatment period 2.5 years of median study drug exposure and 2.8 year of median follow-up
Population: PP (Per Protocol) Analysis set; which included all randomized subjects who received at least 1 dose of randomized study drug and did not have any major protocol violations. The time period included the time the subject was taking study drug and up to 3 days after their last dose (On Treatment Period).
Measure: Number; unit: number of participants with event
Arm/Group | Low Dose Edoxaban/Placebo Warfarin | High Dose Edoxaban/Placebo Warfarin | Warfarin/Placebo Edoxaban
Number analyzed (Participants) | 6982 | 6995 | 6996
number of participants with event | 253 | 182 | 231
Statistical Analysis 1: Comparison: High Dose Edoxaban/Placebo Warfarin vs Warfarin/Placebo Edoxaban; The non-inferiority analysis included the mITT and PP analysis sets for both the on treatment and overall study period, although mITT on-treatment was considered primary; Test type: Non-Inferiority or Equivalence — The primary efficacy endpoint, time to the first occurrence of stroke/SEE, was first compared concurrently between each of the 2 edoxaban groups and warfarin group using the mITT Analysis Set in the on-treatment period for non-inferiority. In order to control the study-wise type-I error rate of two-sided α=0.05 for non-inferiority, each of these 2 comparisons were performed at the statistical significance level of two-sided α=0.025, respectively; p < .0001, Cox proportional hazards model; Hazard Ratio (HR) = 0.79, 97.5% CI 2-sided [.634 to .989]
Statistical Analysis 2: Comparison: Low Dose Edoxaban/Placebo Warfarin vs Warfarin/Placebo Edoxaban; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p = .0064, Cox proportional hazards model; Hazard Ratio (HR) = 1.08, 97.5% CI 2-sided [.878 to 1.32]

4. Primary Outcome: Compare Edoxaban to Warfarin for Composite of Stroke and Systemic Embolic Events (SEE).
Description: The composite of stroke and Systemic Embolic Events (SEE) during the overall study period in the PP (per protocol) analysis set population.
Time Frame: overall study period 2.5 years of median study drug exposure and 2.8 year of median follow-up
Population: PP (per Protocol) Analysis set; which included all randomized subjects who received 1 or more dose of study drug for the overall study period (first dose to end of study) and did not have any major protocol violations. The time period included from the reference date (initial dose of study drug date) to the common study end date (CSED) Visit.
Measure: Number; unit: number of participants with event
Arm/Group | Low Dose Edoxaban/Placebo Warfarin | High Dose Edoxaban/Placebo Warfarin | Warfarin/Placebo Edoxaban
Number analyzed (Participants) | 6982 | 6995 | 6993
number of participants with event | 382 | 292 | 335
Statistical Analysis 1: Comparison: High Dose Edoxaban/Placebo Warfarin vs Warfarin/Placebo Edoxaban; The non-inferiority analysis included the mITT and PP analysis sets for both the on-treatment and overall study period, although mITT on-treatment was considered primary; Test type: Non-Inferiority or Equivalence — In order to control the study-wise type-I error rate of two-sided α=0.05 for non-inferiority, each of these 2 comparisons were performed at the statistical significance level of two-sided α=0.025, respectively. If the upper limit of this CI of the hazard ratio was below 1.38, then non-inferiority to warfarin was considered established for the edoxaban treatment group; p < .0001, Cox proportional hazards model; Hazard Ratio (HR) = .86, 97.5% CI 2-sided [.720 to 1.032]
Statistical Analysis 2: Comparison: Low Dose Edoxaban/Placebo Warfarin vs Warfarin/Placebo Edoxaban; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; p = .0084, Cox proportional hazards model; Hazard Ratio (HR) = 1.13, 97.5% CI 2-sided [.958 to 1.34]

5. Primary Outcome: Compare Edoxaban to Warfarin for Superiority for Composite of Stroke and Systemic Embolic Events (SEE).
Description: Compare edoxaban to warfarin for the composite of stroke and Systemic Embolic Events (SEE) during the overall study period in the ITT analysis set with a superiority analysis.
Time Frame: overall study period 2.5 years of median study drug exposure and 2.8 year of median follow-up
Population: ITT (Intent To Treat) Analysis set; which included all randomized subjects whether or not they received a single dose of randomized study drug. The time frame included from reference date (randomization date) to the common study end date (CSED) Visit.
Measure: Number; unit: number of participants with event
Arm/Group | Low Dose Edoxaban/Placebo Warfarin | High Dose Edoxaban/Placebo Warfarin | Warfarin/Placebo Edoxaban
Number analyzed (Participants) | 7034 | 7035 | 7036
number of participants with event | 383 | 296 | 337
Statistical Analysis 1: Comparison: High Dose Edoxaban/Placebo Warfarin vs Warfarin/Placebo Edoxaban; The superiority analysis included the ITT analysis set; Test type: Superiority or Other; p = .081, Log Rank; Hazard Ratio (HR) = 0.87, 99% CI 2-sided [.709 to 1.068]

6. Secondary Outcome: Compare Edoxaban to Warfarin for Composite of Stroke, Systemic Embolic Event (SEE), and Cardiovascular (CV) Mortality
Description: Compare edoxaban to warfarin for the composite of stroke, Systemic Embolic Events, and Cardiovascular mortality during the overall study period in the ITT analysis set.
Time Frame: overall study period 2.5 years of median study drug exposure and 2.8 year of median follow-up
Population: ITT (Intent To Treat) Analysis set; overall study period, which included all randomized subjects whether or not they received a single dose of randomized study drug. The time frame included from reference date (randomization date) to the common study end date (CSED) Visit..
Measure: Number; unit: number of participants with event
Arm/Group | Low Dose Edoxaban/Placebo Warfarin | High Dose Edoxaban/Placebo Warfarin | Warfarin/Placebo Edoxaban
Number analyzed (Participants) | 7034 | 7035 | 7036
number of participants with event | 796 | 728 | 831
Statistical Analysis 1: Comparison: High Dose Edoxaban/Placebo Warfarin vs Warfarin/Placebo Edoxaban; the time to first event was estimated by a KM estimate and was compared between the edoxaban 60 mg group and the warfarin group using a log-rank test at a pairwise comparison significance level of α=0.01; Test type: Superiority or Other; p = .0053, Log Rank; Hazard Ratio (HR) = .87, 95% CI 2-sided [.786 to .959]

7. Secondary Outcome: Compare Edoxaban to Warfarin for Major Adverse Cardiac Event (MACE): a Composite of Non-fatal MI, Non-fatal Stroke, Non-fatal SEE, and Death Due to CV Cause or Bleeding
Description: Compare edoxaban to warfarin for Major Adverse Cardiac Event (MACE): a composite of non-fatal Myocardial Infarction, non-fatal stroke, non-fatal Systemic Embolic Events, and death due to Cardiovascular cause or bleeding during the overall study period in the ITT analysis set.
Time Frame: overall study period 2.5 years of median study drug exposure and 2.8 year of median follow-up
Population: ITT overall study period, which included all randomized subjects whether or not they received a single dose of randomized study drug. The time frame included from the reference date (randomization date) to the common study end date (CSED) Visit.
Measure: Number; unit: number of participants with event
Arm/Group | Low Dose Edoxaban/Placebo Warfarin | High Dose Edoxaban/Placebo Warfarin | Warfarin/Placebo Edoxaban
Number analyzed (Participants) | 7034 | 7035 | 7036
number of participants with event | 913 | 827 | 926
Statistical Analysis 1: Comparison: High Dose Edoxaban/Placebo Warfarin vs Warfarin/Placebo Edoxaban; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = .0109, Log Rank; Hazard Ratio (HR) = .89, 95% CI 2-sided [.806 to .972]

8. Secondary Outcome: Compare Edoxaban to Warfarin for Composite of Stroke, SEE, and All-cause Mortality
Description: Compare Edoxaban to warfarin for Composite of stroke, Systemic Embolic Events, and all-cause mortality during the overall study period in the ITT analysis set.
Time Frame: overall study period 2.5 years of median study drug exposure and 2.8 year of median follow-up
Population: as for outcome 7
Measure: Number; unit: number of participants with event
Arm/Group | Low Dose Edoxaban/Placebo Warfarin | High Dose Edoxaban/Placebo Warfarin | Warfarin/Placebo Edoxaban
Number analyzed (Participants) | 7034 | 7035 | 7036
number of participants with event | 985 | 949 | 1046
Statistical Analysis 1: Comparison: High Dose Edoxaban/Placebo Warfarin vs Warfarin/Placebo Edoxaban; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = .0168, Log Rank; Hazard Ratio (HR) = .90, 95% CI 2-sided [.823 to .981]

9. Secondary Outcome: Adjudicated Bleeding Events
Description: Compare edoxaban versus warfarin for Adjudicated Bleeding Events during the on-treatment period in the Safety Analysis set.
  Major bleeding was adjudicated by the Clinical Events Committee (CEC) and defined based on published guidance from the International Society on Thrombosis and Haemostasis (ISTH), with minor modifications for Hgb decrease and blood transfusion requirements.
Time Frame: on-treatment period 2.5 years of median study drug exposure and 2.8 year of median follow-up
Population: Safety-analysis set, on-treatment period
Measure: Number; unit: number of participants with event
Arm/Group | Low Dose Edoxaban/Placebo Warfarin | High Dose Edoxaban/Placebo Warfarin | Warfarin/Placebo Edoxaban
Number analyzed (Participants) | 7002 | 7012 | 7012
number of participants with event
  Major bleed | 254 | 418 | 524
  ICH Major bleed | 41 | 61 | 132
  Non-ICH Major bleed | 214 | 359 | 398
  Fatal bleed | 21 | 32 | 59
  non-fatal (Major) bleed | 234 | 386 | 466
  life-threatening bleed | 40 | 62 | 122
  clinically relevant non-major bleed | 969 | 1214 | 1396
  major or clinically relevant non-major | 1161 | 1528 | 1761
  minor | 533 | 604 | 714
  any confirmed bleed | 1499 | 1865 | 2114
Statistical Analysis 1: Comparison: High Dose Edoxaban/Placebo Warfarin vs Warfarin/Placebo Edoxaban; All Major Adjudicated Bleeding Events, Safety Analysis Set On-treatment period; Test type: Superiority or Other; p = .0009, Regression, Cox; Cox Proportional Hazard = .80, 95% CI 2-sided [.707 to .914]
Statistical Analysis 2: Comparison: Low Dose Edoxaban/Placebo Warfarin vs Warfarin/Placebo Edoxaban; All Major Adjudicated Bleeding Events, Safety Analysis Set On-treatment period. The HR, two-sided CI, and p-value for pairwise comparisons versus Warfarin are based on the Cox regression model with counting process approach for on-treatment including treatment and the two stratification factors as covariates: the dichotomized CHADS2 score and the dichotomized dose-adjustment factor; Test type: Superiority or Other; p < .0001, Regression, Cox; Cox Proportional Hazard = 0.47, 95% CI 2-sided [.406 to .548]
Statistical Analysis 3: Comparison: High Dose Edoxaban/Placebo Warfarin vs Warfarin/Placebo Edoxaban; Major or Clinically Relevant Non-Major, high dose vs. warfarin; Test type: Superiority or Other; p < .0001, Regression, Cox; Cox Proportional Hazard = .86, 95% CI 2-sided [.800 to .918]
Statistical Analysis 4: Comparison: Low Dose Edoxaban/Placebo Warfarin vs Warfarin/Placebo Edoxaban; Major or Clinically Relevant Non-Major, low dose vs. warfarin; Test type: Superiority or Other; p < .0001, Regression, Cox; Cox Proportional Hazard = .62, 95% CI 2-sided [.575 to .666]

ADVERSE EVENTS:
Time Frame: On treatment (safety analysis set)
Groups:
- High Dose Edoxaban/Placebo Warfarin: Edoxaban tablets plus warfarin placebo tablets
  Edoxaban tablets (high dose regimen): Edoxaban tablets plus warfarin placebo tablets each taken once daily for 24 months
  placebo warfarin: placebo warfarin
- Low Dose Edoxaban/Placebo Warfarin: Edoxaban tablets plus warfarin placebo tablets
  Edoxaban tablets (low dose regimen): Edoxaban tablets plus warfarin placebo tablets each taken once daily for 24 months
  placebo warfarin: placebo warfarin
Arm/Group | Warfarin/Placebo Edoxaban | High Dose Edoxaban/Placebo Warfarin | Low Dose Edoxaban/Placebo Warfarin
Serious Adverse Events (participants affected / at risk) | 3581/7012 | 3393/7012 | 3448/7002
Other Adverse Events (participants affected / at risk) | 4200/7012 | 4201/7012 | 4057/7002
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Warfarin/Placebo Edoxaban (N=7012) | High Dose Edoxaban/Placebo Warfarin (N=7012) | Low Dose Edoxaban/Placebo Warfarin (N=7002)
PNEUMONIA (Infections and infestations) | 262 (292) | 259 (298) | 219 (237)
URINARY TRACT INFECTION (Infections and infestations) | 78 (86) | 60 (75) | 57 (62)
BRONCHITIS (Infections and infestations) | 60 (64) | 56 (58) | 57 (63)
CELLULITIS (Infections and infestations) | 62 (71) | 52 (64) | 59 (69)
SEPSIS (Infections and infestations) | 35 (35) | 38 (39) | 43 (44)
GASTROENTERITIS (Infections and infestations) | 30 (31) | 27 (29) | 29 (29)
LOBAR PNEUMONIA (Infections and infestations) | 24 (25) | 23 (24) | 23 (23)
BRONCHOPNEUMONIA (Infections and infestations) | 35 (35) | 22 (24) | 29 (29)
DIVERTICULITIS (Infections and infestations) | 22 (26) | 15 (15) | 10 (10)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 8 (8) | 15 (17) | 14 (14)
SEPTIC SHOCK (Infections and infestations) | 27 (27) | 14 (14) | 16 (16)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 7 (8) | 12 (12) | 10 (10)
ERYSIPELAS (Infections and infestations) | 15 (19) | 11 (12) | 19 (19)
OSTEOMYELITIS (Infections and infestations) | 11 (12) | 10 (10) | 13 (16)
PNEUMONIA BACTERIAL (Infections and infestations) | 14 (15) | 10 (11) | 11 (13)
APPENDICITIS (Infections and infestations) | 9 (9) | 9 (9) | 8 (8)
PYELONEPHRITIS (Infections and infestations) | 13 (17) | 9 (9) | 5 (5)
UROSEPSIS (Infections and infestations) | 13 (13) | 9 (10) | 19 (22)
CYSTITIS (Infections and infestations) | 2 (2) | 8 (8) | 1 (1)
PYELONEPHRITIS ACUTE (Infections and infestations) | 5 (5) | 8 (8) | 3 (3)
GASTROENTERITIS VIRAL (Infections and infestations) | 6 (6) | 7 (8) | 3 (3)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 6 (7) | 7 (7) | 3 (3)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 2 (2) | 6 (8) | 3 (3)
GANGRENE (Infections and infestations) | 9 (9) | 6 (7) | 8 (10)
INFECTION (Infections and infestations) | 2 (2) | 6 (6) | 6 (6)
INFLUENZA (Infections and infestations) | 5 (5) | 6 (6) | 6 (6)
LUNG INFECTION (Infections and infestations) | 6 (7) | 6 (7) | 3 (3)
CHOLECYSTITIS INFECTIVE (Infections and infestations) | 2 (2) | 5 (5) | 3 (3)
HERPES ZOSTER (Infections and infestations) | 4 (4) | 5 (6) | 9 (9)
INFECTED SKIN ULCER (Infections and infestations) | 2 (2) | 5 (5) | 5 (5)
INFECTIOUS PERITONITIS (Infections and infestations) | 2 (2) | 5 (5) | 4 (4)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 9 (9) | 5 (6) | 8 (8)
ENDOCARDITIS (Infections and infestations) | 5 (5) | 4 (4) | 6 (6)
ORCHITIS (Infections and infestations) | 1 (1) | 4 (5) | 4 (4)
PULMONARY TUBERCULOSIS (Infections and infestations) | 1 (1) | 4 (4) | 2 (2)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 2 (2) | 4 (4) | 1 (1)
WOUND INFECTION (Infections and infestations) | 5 (5) | 4 (4) | 3 (3)
ABSCESS LIMB (Infections and infestations) | 4 (4) | 3 (3) | 4 (4)
BACTERIAL SEPSIS (Infections and infestations) | 0 (0) | 3 (3) | 2 (2)
CLOSTRIDIAL INFECTION (Infections and infestations) | 0 (0) | 3 (4) | 2 (2)
GASTROENTERITIS SALMONELLA (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
IMPLANT SITE INFECTION (Infections and infestations) | 3 (3) | 3 (3) | 1 (1)
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 0 (0) | 3 (3) | 4 (4)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 2 (2) | 3 (3) | 2 (2)
TRACHEOBRONCHITIS (Infections and infestations) | 3 (3) | 3 (3) | 2 (2)
URINARY TRACT INFECTION PSEUDOMONAL (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
VIRAL INFECTION (Infections and infestations) | 3 (3) | 3 (3) | 6 (6)
APPENDICITIS PERFORATED (Infections and infestations) | 2 (2) | 2 (2) | 2 (2)
ARTHRITIS BACTERIAL (Infections and infestations) | 8 (8) | 2 (2) | 3 (3)
BACTERAEMIA (Infections and infestations) | 2 (2) | 2 (2) | 2 (2)
BRONCHITIS BACTERIAL (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
CAMPYLOBACTER GASTROENTERITIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
CREUTZFELDT-JAKOB DISEASE (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 2 (2) | 2 (2) | 4 (5)
DIABETIC GANGRENE (Infections and infestations) | 5 (5) | 2 (4) | 3 (3)
DIARRHOEA INFECTIOUS (Infections and infestations) | 1 (1) | 2 (2) | 2 (2)
ENDOCARDITIS BACTERIAL (Infections and infestations) | 2 (2) | 2 (2) | 2 (2)
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
ESCHERICHIA SEPSIS (Infections and infestations) | 3 (3) | 2 (2) | 2 (2)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 6 (6) | 2 (2) | 2 (2)
HEPATITIS E (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
INTERVERTEBRAL DISCITIS (Infections and infestations) | 2 (2) | 2 (2) | 3 (3)
KLEBSIELLA BACTERAEMIA (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
LARYNGITIS (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
LOCALISED INFECTION (Infections and infestations) | 4 (4) | 2 (2) | 3 (3)
LUNG INFECTION PSEUDOMONAL (Infections and infestations) | 0 (0) | 2 (2) | 4 (4)
NECROTISING FASCIITIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
PERIORBITAL CELLULITIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
PERITONITIS BACTERIAL (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 2 (2) | 2 (2) | 2 (2)
PULMONARY SEPSIS (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
SALMONELLOSIS (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
SCROTAL ABSCESS (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
SINUSITIS (Infections and infestations) | 2 (2) | 2 (2) | 3 (3)
SOFT TISSUE INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 10 (11) | 2 (2) | 7 (7)
STREPTOCOCCAL SEPSIS (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
TOOTH ABSCESS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
TUBERCULOUS PLEURISY (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
URINARY TRACT INFECTION BACTERIAL (Infections and infestations) | 4 (5) | 2 (2) | 2 (2)
WOUND INFECTION STAPHYLOCOCCAL (Infections and infestations) | 1 (1) | 2 (2) | 2 (2)
ABDOMINAL ABSCESS (Infections and infestations) | 2 (2) | 1 (1) | 2 (2)
ABDOMINAL WALL ABSCESS (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ABSCESS INTESTINAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ACINETOBACTER BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
AMOEBIC COLITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ANAL ABSCESS (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
ARTERIOSCLEROTIC GANGRENE (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ARTHRITIS INFECTIVE (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
ATYPICAL MYCOBACTERIAL PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
BACTERIAL PROSTATITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
BACTEROIDES BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
BILIARY SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
BRAIN ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
BRONCHIOLITIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
CANDIDA PNEUMONIA (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
CELLULITIS STAPHYLOCOCCAL (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
CHOLANGITIS SUPPURATIVE (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CYSTITIS KLEBSIELLA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
DENGUE FEVER (Infections and infestations) | 0 (0) | 1 (1) | 4 (4)
DEVICE RELATED SEPSIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
DISSEMINATED TUBERCULOSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ECZEMA INFECTED (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
EMPYEMA (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
ENCEPHALITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ENTEROCOCCAL BACTERAEMIA (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
ENTEROCOCCAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
ENTEROCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 1 (2) | 1 (1)
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
ESCHERICHIA INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
FEBRILE INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
FURUNCLE (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
GAS GANGRENE (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
GASTRIC ULCER HELICOBACTER (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
GASTRITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
GASTROENTERITIS AEROMONAS (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
GROIN ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 4 (4)
HAEMATOMA INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
HELICOBACTER GASTRITIS (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
HEPATIC CYST INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
HEPATITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
HERPES ZOSTER OPHTHALMIC (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
INFECTIOUS PLEURAL EFFUSION (Infections and infestations) | 3 (4) | 1 (1) | 0 (0)
INFECTIVE MYOSITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
INFUSION SITE INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
KLEBSIELLA SEPSIS (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
LABYRINTHITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION BACTERIAL (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
LYMPH NODE TUBERCULOSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
MASTOIDITIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
MENINGITIS MENINGOCOCCAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
MYIASIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
NEUROCYSTICERCOSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
NEUTROPENIC SEPSIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
NOSOCOMIAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
PARAOESOPHAGEAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PERITONSILLAR ABSCESS (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
PHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
PNEUMONIA HAEMOPHILUS (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
PNEUMONIA NECROTISING (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA PRIMARY ATYPICAL (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
PNEUMONIA VIRAL (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
POST PROCEDURAL CELLULITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PSEUDOMEMBRANOUS COLITIS (Infections and infestations) | 0 (0) | 1 (1) | 2 (3)
PSEUDOMONAL BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PSEUDOMONAS BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PULMONARY TUBERCULOMA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PYELONEPHRITIS CHRONIC (Infections and infestations) | 2 (3) | 1 (1) | 3 (3)
SEPSIS SYNDROME (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
SEPTIC ARTHRITIS STAPHYLOCOCCAL (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
SIALOADENITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
SINOBRONCHITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
SKIN INFECTION (Infections and infestations) | 1 (1) | 1 (2) | 1 (1)
STAPHYLOCOCCAL SKIN INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
STREPTOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
SUBDIAPHRAGMATIC ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
TOXIC SHOCK SYNDROME (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
VESTIBULAR NEURONITIS (Infections and infestations) | 5 (5) | 1 (1) | 0 (0)
VIRAL DIARRHOEA (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
VIRAL LABYRINTHITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
VIRAL PHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
WOUND SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL SEPSIS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
ABSCESS ORAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ACARODERMATITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
ACINETOBACTER INFECTION (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
AMERICAN TRYPANOSOMIASIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
BACTERIAL FOOD POISONING (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
BRONCHITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
BURSITIS INFECTIVE (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
CAMPYLOBACTER INTESTINAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
CARBUNCLE (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
CELLULITIS GANGRENOUS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
CELLULITIS STREPTOCOCCAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
CHIKUNGUNYA VIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
CHRONIC SINUSITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
CHRONIC TONSILLITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
CITROBACTER SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
CYSTITIS BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
CYSTITIS ESCHERICHIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
DIABETIC FOOT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
DOUGLAS' ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
EMPHYSEMATOUS CHOLECYSTITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ENCEPHALITIS HERPES (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ENDOCARDITIS ENTEROCOCCAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ENTERITIS INFECTIOUS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ENTEROBACTER BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ENTEROBACTER SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
EPIGLOTTITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
EXTRADURAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
GASTROENTERITIS BACTERIAL (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
GASTROENTERITIS CLOSTRIDIAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
GASTROENTERITIS ROTAVIRUS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
GASTROINTESTINAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
GINGIVAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
GROIN INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
H1N1 INFLUENZA (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
HAEMOPHILUS INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
HELICOBACTER INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
HEPATITIS B (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
HEPATITIS INFECTIOUS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
IMPLANT SITE ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
INCISION SITE INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
INFECTED DERMAL CYST (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
JOINT ABSCESS (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
KERATITIS HERPETIC (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
KIDNEY INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
LEGIONELLA INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
LIVER ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
LOWER RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
MALARIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
MENINGITIS ASEPTIC (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
MENINGITIS BACTERIAL (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
MENINGITIS STREPTOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
MENINGITIS TUBERCULOUS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
MENINGITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
MOLLUSCUM CONTAGIOSUM (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
MURINE TYPHUS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
MUSCLE ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
MYCOTOXICOSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
NEUROBORRELIOSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
OSTEOMYELITIS CHRONIC (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
OTITIS MEDIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTITIS MEDIA ACUTE (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PARONYCHIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PAROTITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PERICORONITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PERIRECTAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PLASMODIUM FALCIPARUM INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA FUNGAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA INFLUENZAL (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
PNEUMONIA KLEBSIELLA (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
PNEUMONIA LEGIONELLA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA MYCOPLASMAL (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
POST PROCEDURAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
POST PROCEDURAL PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PROTEUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PSEUDOMONAS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
PSOAS ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
RECTAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
RENAL CYST INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
RETROPERITONEAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
SEPTIC ARTHRITIS STREPTOCOCCAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
SEPTIC EMBOLUS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
SEPTIC ENCEPHALOPATHY (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
SERRATIA SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
SPLENIC ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
STREPTOCOCCAL BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
TUBERCULOSIS OF CENTRAL NERVOUS SYSTEM (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
TYPHOID FEVER (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
URINARY TRACT INFECTION ENTEROCOCCAL (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
VULVAL CELLULITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 32 (32) | 34 (34) | 34 (34)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 37 (38) | 29 (29) | 30 (30)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 23 (23) | 21 (31) | 26 (36)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 (18) | 18 (18) | 19 (19)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 (15) | 16 (16) | 13 (13)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (10) | 13 (13) | 4 (5)
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 (15) | 10 (10) | 12 (12)
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 9 (9) | 6 (6)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 9 (9) | 6 (6)
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 9 (9) | 7 (7)
BLADDER TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (12) | 8 (8) | 13 (13)
PROSTATIC ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 8 (8) | 2 (2)
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 7 (7) | 1 (1)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (11) | 7 (7) | 4 (19)
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (9) | 6 (6) | 8 (8)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 6 (6) | 6 (6)
UTERINE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 6 (6) | 2 (2)
BRONCHIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 5 (5) | 0 (0)
ADENOCARCINOMA PANCREAS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4) | 4 (4)
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4) | 1 (1)
OESOPHAGEAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4) | 3 (3)
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4) | 8 (8)
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 4 (4) | 7 (7)
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4) | 1 (1)
SMALL CELL LUNG CANCER STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4) | 3 (3)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 4 (4) | 8 (10)
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 4 (4) | 5 (5)
COLORECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3) | 3 (3)
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3) | 4 (4)
GASTRIC CANCER STAGE 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 3 (3) | 1 (1)
GASTROINTESTINAL STROMAL TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 0 (0)
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 2 (2)
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3) | 0 (0)
LUNG SQUAMOUS CELL CARCINOMA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3) | 5 (5)
OESOPHAGEAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 0 (0)
PANCREATIC CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3) | 4 (4)
PROSTATE CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3) | 1 (1)
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 3 (3) | 4 (4)
THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3) | 1 (1)
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2) | 3 (3)
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1)
BILE DUCT CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 3 (3)
BLADDER CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2) | 1 (1)
BRAIN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 3 (3)
DIFFUSE LARGE B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2) | 1 (1)
FIBROADENOMA OF BREAST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
GALLBLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 2 (2)
GASTRIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1)
GASTROINTESTINAL TRACT ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0)
LARYNGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2) | 2 (2)
LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
LUNG ADENOCARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 2 (2) | 1 (1)
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 1 (1)
MENINGIOMA BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 3 (3)
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 2 (2) | 3 (3)
METASTATIC GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 2 (2)
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 3 (3)
OVARIAN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2) | 1 (1)
PANCREATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0)
PARATHYROID TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
PLASMACYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2) | 3 (3)
URETERIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 2 (2)
ABDOMINAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
ACUTE PROMYELOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
ANGIOSARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
BENIGN DUODENAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
BENIGN GASTRIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
BENIGN LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 2 (2)
BENIGN NEOPLASM OF ADRENAL GLAND (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
BENIGN NEOPLASM OF BLADDER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
BENIGN NEOPLASM OF PROSTATE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
BENIGN NEOPLASM OF URETHRA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
BENIGN PANCREATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
BENIGN SALIVARY GLAND NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 1 (1)
BENIGN URINARY TRACT NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
BILIARY NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
BLADDER NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 1 (1)
BONE CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
BONE GIANT CELL TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
BREAST CANCER STAGE II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
BREAST NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
BRONCHIAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
COLON CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
FOLLICLE CENTRE LYMPHOMA, FOLLICULAR GRADE I, II, III STAGE III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
GASTRIC CANCER STAGE II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
GLIOBLASTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
HAEMANGIOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
HEAD AND NECK CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
HEPATIC CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 1 (1) | 1 (1)
HEPATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
HODGKIN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
HYPOPHARYNGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
INTRADUCTAL PAPILLOMA OF BREAST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
IRITIC MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
KERATOACANTHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
LARGE INTESTINE CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
LARYNGEAL PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
LIP AND/OR ORAL CAVITY CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
LUNG ADENOCARCINOMA STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
LUNG CARCINOMA CELL TYPE UNSPECIFIED STAGE III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 4 (4)
LYMPHANGIOSIS CARCINOMATOSA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
LYMPHOPLASMACYTOID LYMPHOMA/IMMUNOCYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
MALIGNANT NEOPLASM OF PLEURA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
MALIGNANT PALATE NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2)
MANTLE CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
MELANOMA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
MENINGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
MESOTHELIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 2 (2)
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 3 (3)
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
METASTATIC BRONCHIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
METASTATIC MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 1 (1) | 0 (0)
METASTATIC PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
METASTATIC SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 2 (2)
NEOPLASM PROSTATE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
NEUROENDOCRINE TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
NON-HODGKIN'S LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1) | 1 (1)
NON-HODGKIN'S LYMPHOMA STAGE I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 2 (2)
NON-SMALL CELL LUNG CANCER STAGE I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
OESOPHAGEAL ADENOCARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
OESOPHAGEAL ADENOCARCINOMA STAGE II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
OESOPHAGEAL SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
ORAL PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
OVARIAN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
PARANEOPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
PARATHYROID TUMOUR MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
PHARYNGEAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
RECTAL CANCER STAGE I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
RECTOSIGMOID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
RENAL ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
SEBORRHOEIC KERATOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
SINONASAL PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
SMALL INTESTINE CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
THYROID ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 2 (2)
URINARY TRACT NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
ACUTE LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
ADRENAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
ANGIOSARCOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
BENIGN BILIARY NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
BENIGN BREAST NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1)
BENIGN COLONIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (3)
BENIGN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2)
BENIGN NEOPLASM OF CERVIX UTERI (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
BENIGN NEOPLASM OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
BENIGN NEOPLASM OF THYROID GLAND (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
BENIGN PENILE NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
BENIGN RENAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
BLADDER PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
BLADDER TRANSITIONAL CELL CARCINOMA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
BONE NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
BONE NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
BOWEN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
BRAIN NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
BREAST CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 2 (2)
BREAST CANCER STAGE I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
BRONCHIOLOALVEOLAR CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
CARCINOID TUMOUR OF THE DUODENUM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
CARCINOID TUMOUR PULMONARY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
CARDIAC MYXOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
CENTRAL NERVOUS SYSTEM LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
CEREBELLAR TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
CERVIX CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
CHOLESTEATOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
CHRONIC LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 3 (3)
CHRONIC MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
COLON CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
COLON CANCER STAGE II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
COLON NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 3 (3)
ESSENTIAL THROMBOCYTHAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
FOLLICLE CENTRE LYMPHOMA, FOLLICULAR GRADE I, II, III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
FOLLICLE CENTRE LYMPHOMA, FOLLICULAR GRADE I, II, III STAGE II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
GASTRIC ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
GENITOURINARY TRACT NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
GLIOBLASTOMA MULTIFORME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
GLIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
HAEMANGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
INTESTINAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2)
LARGE CELL CARCINOMA OF THE RESPIRATORY TRACT STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
LARYNGEAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
LENTIGO MALIGNA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
LUNG CARCINOMA CELL TYPE UNSPECIFIED STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
LUNG INFILTRATION MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
LUNG SQUAMOUS CELL CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
LUNG SQUAMOUS CELL CARCINOMA STAGE I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
LUNG SQUAMOUS CELL CARCINOMA STAGE III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
LYMPHOCYTIC LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
MALIGNANT ASCITES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
MALIGNANT MELANOMA IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
MALIGNANT MESENCHYMOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
MALIGNANT NEOPLASM OF AMPULLA OF VATER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
MALIGNANT NEOPLASM OF RENAL PELVIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
MALIGNANT PERITONEAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
METASTASES TO GALLBLADDER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
METASTASES TO LARGE INTESTINE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
METASTASES TO LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 2 (2)
METASTASES TO PERITONEUM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
METASTASES TO SPINE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
METASTATIC LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
MULTIPLE MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 0 (0) | 3 (3)
NASAL CAVITY CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
NASOPHARYNGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
NEOPLASM SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
NEUROENDOCRINE CARCINOMA OF THE SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
NON-SMALL CELL LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
OVARIAN ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
PENIS CARCINOMA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
PITUITARY TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2)
RECTAL ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
RECTAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
REFRACTORY CYTOPENIA WITH MULTILINEAGE DYSPLASIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
RENAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2)
RENAL CANCER STAGE II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
RENAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
RENAL ONCOCYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
RETROPERITONEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
SALIVARY GLAND ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
SARCOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
SMALL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
SPINAL HAEMANGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
TESTIS CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
TONGUE NEOPLASM MALIGNANT STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
TONSIL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
UNDIFFERENTIATED SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
URETERAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
URETHRAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
UTERINE LEIOMYOSARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
VULVAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
VULVAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
VULVAL CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
ANAEMIA (Blood and lymphatic system disorders) | 62 (74) | 91 (106) | 70 (77)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 13 (14) | 34 (37) | 14 (15)
SPONTANEOUS HAEMATOMA (Blood and lymphatic system disorders) | 22 (23) | 10 (10) | 5 (5)
HYPOCHROMIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 6 (6) | 2 (2)
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 4 (4) | 3 (3) | 8 (8)
NORMOCHROMIC NORMOCYTIC ANAEMIA (Blood and lymphatic system disorders) | 5 (5) | 3 (3) | 3 (13)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 1 (2)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2)
LYMPHADENITIS (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1)
MICROCYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 3 (3)
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 3 (3)
ANAEMIA MEGALOBLASTIC (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
ANAEMIA OF CHRONIC DISEASE (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
ANAEMIA VITAMIN B12 DEFICIENCY (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
AUTOIMMUNE THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
COAGULOPATHY (Blood and lymphatic system disorders) | 9 (10) | 1 (1) | 4 (4)
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2)
HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
MACROCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
POLYCYTHAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
THROMBOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
ANAEMIA FOLATE DEFICIENCY (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
ANAEMIA MACROCYTIC (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
ANAEMIA OF MALIGNANT DISEASE (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 3 (3)
APLASTIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
BONE MARROW FAILURE (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
HAEMORRHAGIC DIATHESIS (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
HEPARIN-INDUCED THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERCOAGULATION (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
HYPOCOAGULABLE STATE (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
IDIOPATHIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
LYMPHADENOPATHY MEDIASTINAL (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
NEPHROGENIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
PERNICIOUS ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
SPLENOMEGALY (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
DRUG HYPERSENSITIVITY (Immune system disorders) | 3 (3) | 3 (3) | 1 (1)
HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 2 (2) | 2 (2)
ANAPHYLACTIC REACTION (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
ANAPHYLACTIC SHOCK (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
SECONDARY IMMUNODEFICIENCY (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
ALLERGY TO ARTHROPOD BITE (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
AMYLOIDOSIS (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
SARCOIDOSIS (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
GOITRE (Endocrine disorders) | 1 (1) | 3 (3) | 6 (6)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1) | 3 (3) | 0 (0)
HYPERTHYROIDISM (Endocrine disorders) | 5 (5) | 2 (3) | 6 (6)
CARCINOID SYNDROME (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERPARATHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
INAPPROPRIATE ANTIDIURETIC HORMONE SECRETION (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
AUTOIMMUNE THYROIDITIS (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
BASEDOW'S DISEASE (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERPARATHYROIDISM PRIMARY (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
MYXOEDEMA (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
SECONDARY ADRENOCORTICAL INSUFFICIENCY (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
THYROIDITIS (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 33 (33) | 28 (31) | 42 (45)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 16 (18) | 24 (24) | 16 (17)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 18 (18) | 21 (21) | 36 (41)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 16 (17) | 15 (15) | 13 (13)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 (2) | 11 (11) | 9 (10)
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 7 (7) | 10 (10) | 15 (18)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 3 (3) | 7 (7) | 15 (17)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 11 (11) | 6 (6) | 8 (10)
GOUT (Metabolism and nutrition disorders) | 4 (4) | 5 (5) | 4 (4)
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 4 (4) | 5 (5) | 5 (5)
DIABETIC FOOT (Metabolism and nutrition disorders) | 10 (10) | 4 (4) | 3 (4)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 3 (3)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (3)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1)
FLUID OVERLOAD (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 0 (0)
MALNUTRITION (Metabolism and nutrition disorders) | 2 (3) | 2 (2) | 1 (1)
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
CACHEXIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
HYPEROSMOLAR STATE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERVOLAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 4 (4)
METABOLIC DISORDER (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
SHOCK HYPOGLYCAEMIC (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
CALCIPHYLAXIS (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3)
FOLATE DEFICIENCY (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
IRON DEFICIENCY (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
LACTIC ACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
NEUROGLYCOPENIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
OBESITY (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
VITAMIN B12 DEFICIENCY (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2)
MENTAL STATUS CHANGES (Psychiatric disorders) | 7 (7) | 12 (13) | 8 (8)
DEPRESSION (Psychiatric disorders) | 5 (5) | 11 (12) | 12 (12)
ANXIETY (Psychiatric disorders) | 4 (4) | 8 (9) | 0 (0)
DELIRIUM (Psychiatric disorders) | 2 (2) | 8 (9) | 4 (5)
CONFUSIONAL STATE (Psychiatric disorders) | 6 (7) | 6 (6) | 5 (5)
ALCOHOL ABUSE (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0)
COMPLETED SUICIDE (Psychiatric disorders) | 2 (2) | 3 (3) | 1 (1)
PSYCHOTIC DISORDER (Psychiatric disorders) | 0 (0) | 3 (3) | 1 (1)
ANXIETY DISORDER (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
SUICIDE ATTEMPT (Psychiatric disorders) | 4 (4) | 2 (2) | 1 (1)
AGITATION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
ALCOHOLISM (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
DEPRESSED MOOD (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
EMOTIONAL DISTRESS (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
HALLUCINATION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
INTENTIONAL SELF-INJURY (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
MENTAL DISORDER (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
ACUTE PSYCHOSIS (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
ACUTE STRESS DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
AGGRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
BIPOLAR DISORDER (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
BURNOUT SYNDROME (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
DELIRIUM TREMENS (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0)
DEPRESSION SUICIDAL (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
DISORIENTATION (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
DRUG ABUSE (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
DRUG DEPENDENCE (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
DYSPHORIA (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
GENERALISED ANXIETY DISORDER (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
MAJOR DEPRESSION (Psychiatric disorders) | 2 (2) | 0 (0) | 3 (3)
MENTAL DISORDER DUE TO A GENERAL MEDICAL CONDITION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
PANIC ATTACK (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
PANIC DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
PSYCHOSOMATIC DISEASE (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
SCHIZOPHRENIA (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 88 (94) | 104 (111) | 125 (138)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 74 (81) | 85 (97) | 107 (125)
ISCHAEMIC STROKE (Nervous system disorders) | 95 (105) | 83 (85) | 141 (152)
SYNCOPE (Nervous system disorders) | 65 (68) | 53 (55) | 64 (65)
CEREBRAL INFARCTION (Nervous system disorders) | 21 (22) | 30 (33) | 45 (51)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 32 (33) | 23 (23) | 11 (11)
DIZZINESS (Nervous system disorders) | 12 (13) | 15 (15) | 15 (17)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 36 (37) | 13 (14) | 12 (12)
CAROTID ARTERY STENOSIS (Nervous system disorders) | 13 (13) | 12 (12) | 12 (12)
PRESYNCOPE (Nervous system disorders) | 10 (10) | 12 (12) | 15 (15)
CONVULSION (Nervous system disorders) | 12 (12) | 11 (12) | 12 (14)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 17 (17) | 11 (13) | 3 (3)
DEMENTIA (Nervous system disorders) | 10 (10) | 8 (8) | 1 (1)
HAEMORRHAGIC STROKE (Nervous system disorders) | 20 (22) | 8 (8) | 6 (7)
GRAND MAL CONVULSION (Nervous system disorders) | 2 (2) | 5 (5) | 5 (5)
VERTEBROBASILAR INSUFFICIENCY (Nervous system disorders) | 10 (12) | 5 (6) | 4 (5)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 6 (6) | 4 (5) | 4 (4)
EMBOLIC STROKE (Nervous system disorders) | 8 (9) | 4 (4) | 5 (5)
EPILEPSY (Nervous system disorders) | 14 (16) | 4 (10) | 14 (15)
HEADACHE (Nervous system disorders) | 5 (5) | 4 (4) | 3 (3)
HEMIPARESIS (Nervous system disorders) | 2 (2) | 4 (4) | 1 (1)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 7 (7) | 4 (4) | 1 (1)
VASCULAR ENCEPHALOPATHY (Nervous system disorders) | 4 (4) | 4 (5) | 5 (5)
BRAIN STEM INFARCTION (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0)
COMPLEX PARTIAL SEIZURES (Nervous system disorders) | 0 (0) | 3 (3) | 2 (2)
DEMENTIA ALZHEIMER'S TYPE (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1)
HYPOXIC-ISCHAEMIC ENCEPHALOPATHY (Nervous system disorders) | 2 (2) | 3 (3) | 2 (2)
LACUNAR INFARCTION (Nervous system disorders) | 7 (7) | 3 (3) | 6 (8)
RADICULOPATHY (Nervous system disorders) | 0 (0) | 3 (3) | 1 (2)
THALAMUS HAEMORRHAGE (Nervous system disorders) | 2 (2) | 3 (3) | 2 (2)
AMNESIA (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
BRAIN STEM HAEMORRHAGE (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1)
BRAIN STEM STROKE (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
CAROTID ARTERY DISEASE (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
CEREBELLAR HAEMORRHAGE (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
CEREBELLAR INFARCTION (Nervous system disorders) | 6 (6) | 2 (2) | 4 (4)
CEREBRAL ARTERIOSCLEROSIS (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2)
CEREBROVASCULAR DISORDER (Nervous system disorders) | 3 (3) | 2 (2) | 3 (3)
DIABETIC NEUROPATHY (Nervous system disorders) | 3 (3) | 2 (2) | 1 (1)
ENCEPHALOPATHY (Nervous system disorders) | 5 (7) | 2 (2) | 2 (2)
INTERCOSTAL NEURALGIA (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0)
PARKINSONISM (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2)
PERIPHERAL SENSORIMOTOR NEUROPATHY (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
SCIATICA (Nervous system disorders) | 5 (5) | 2 (2) | 4 (4)
THROMBOTIC CEREBRAL INFARCTION (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
TRANSIENT GLOBAL AMNESIA (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
VIITH NERVE PARALYSIS (Nervous system disorders) | 2 (2) | 2 (2) | 3 (3)
AMNESTIC DISORDER (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
AMYOTROPHIC LATERAL SCLEROSIS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
APHASIA (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
ASTERIXIS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
ATAXIA (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
BASILAR ARTERY THROMBOSIS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
BRAIN INJURY (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3)
BRAIN MASS (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
BRAIN STEM ISCHAEMIA (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
CAROTID ARTERY OCCLUSION (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
CAROTID SINUS SYNDROME (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 3 (4) | 1 (1) | 2 (2)
CENTRAL NERVOUS SYSTEM LESION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
CEREBELLAR ATAXIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
CEREBRAL ARTERY OCCLUSION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
CEREBRAL ATROPHY (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
CEREBRAL CIRCULATORY FAILURE (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3)
CEREBRAL HAEMATOMA (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
CERVICOBRACHIAL SYNDROME (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
CLUSTER HEADACHE (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
COGNITIVE DISORDER (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
COMA (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
COMA HEPATIC (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
DRUG WITHDRAWAL CONVULSIONS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
DYSARTHRIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
ENCEPHALOMALACIA (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
FACIAL PARESIS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 1 (3) | 0 (0)
HYPERTENSIVE ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 1 (1) | 4 (4)
HYPOAESTHESIA (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
HYPOGLYCAEMIC COMA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
MIGRAINE WITH AURA (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
MONONEUROPATHY MULTIPLEX (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
MOTOR NEURONE DISEASE (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
MYELOPATHY (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
NARCOLEPSY (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
NERVE COMPRESSION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
NEURALGIA (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
NEURITIS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
PARKINSON'S DISEASE (Nervous system disorders) | 3 (4) | 1 (1) | 3 (4)
PARTIAL SEIZURES (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
PARTIAL SEIZURES WITH SECONDARY GENERALISATION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
PUTAMEN HAEMORRHAGE (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
RADICULAR PAIN (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
RADICULAR SYNDROME (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
RADICULITIS LUMBOSACRAL (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
SPINAL CORD DISORDER (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
THROMBOTIC STROKE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
TRIGEMINAL NEURALGIA (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0)
ULNAR NERVE PALSY (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
UNRESPONSIVE TO STIMULI (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
VASCULAR DEMENTIA (Nervous system disorders) | 4 (4) | 1 (1) | 0 (0)
VERTIGO CNS ORIGIN (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
ACOUSTIC NEURITIS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
AKINESIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
ALCOHOL INDUCED PERSISTING DEMENTIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
BALANCE DISORDER (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
BASAL GANGLIA HAEMORRHAGE (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
BRACHIAL PLEXOPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
BRAIN OEDEMA (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
CAROTID ARTERIOSCLEROSIS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
CAROTID ARTERY THROMBOSIS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
CAUDA EQUINA SYNDROME (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
CEREBELLAR ISCHAEMIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
CEREBELLAR SYNDROME (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
CEREBRAL AMYLOID ANGIOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
CEREBRAL ARTERY EMBOLISM (Nervous system disorders) | 3 (3) | 0 (0) | 3 (3)
CEREBRAL HYPOPERFUSION (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
CEREBRAL THROMBOSIS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
CEREBROVASCULAR INSUFFICIENCY (Nervous system disorders) | 3 (3) | 0 (0) | 3 (3)
CERVICAL CORD COMPRESSION (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
CERVICAL MYELOPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
CRITICAL ILLNESS POLYNEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
CUBITAL TUNNEL SYNDROME (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
DEMENTIA WITH LEWY BODIES (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
DEMYELINATING POLYNEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
EMBOLIC CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
ENCEPHALITIS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
ESSENTIAL TREMOR (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
GUILLAIN-BARRE SYNDROME (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
HAEMORRHAGIC CEREBRAL INFARCTION (Nervous system disorders) | 2 (2) | 0 (0) | 3 (3)
HAEMORRHAGIC TRANSFORMATION STROKE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
HYDROCEPHALUS (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
HYPERCAPNIC ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOKINESIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
HYPONATRAEMIC ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
IIIRD NERVE PARALYSIS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
INTRACRANIAL ANEURYSM (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
INTRACRANIAL HAEMATOMA (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
INTRAVENTRICULAR HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
ISCHAEMIC CEREBRAL INFARCTION (Nervous system disorders) | 3 (3) | 0 (0) | 5 (5)
ISCHAEMIC NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
LATERAL MEDULLARY SYNDROME (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
LUMBAR RADICULOPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
MIGRAINE (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
MONOPARESIS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
MYASTHENIA GRAVIS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
NEUROLOGICAL SYMPTOM (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
NEUROMYOPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
NORMAL PRESSURE HYDROCEPHALUS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OPTIC NEURITIS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
ORTHOSTATIC INTOLERANCE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
PARAPLEGIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
PHRENIC NERVE PARALYSIS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
POLYNEUROPATHY (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
POST-TRAUMATIC EPILEPSY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
REVERSIBLE ISCHAEMIC NEUROLOGICAL DEFICIT (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SENILE DEMENTIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SIMPLE PARTIAL SEIZURES (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
SPEECH DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SPINAL HAEMATOMA (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
STATUS EPILEPTICUS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3)
SUBDURAL HYGROMA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
TENSION HEADACHE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
TREMOR (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
VOCAL CORD PARALYSIS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
CATARACT (Eye disorders) | 47 (63) | 58 (65) | 60 (72)
GLAUCOMA (Eye disorders) | 2 (2) | 5 (5) | 4 (5)
VITREOUS HAEMORRHAGE (Eye disorders) | 1 (1) | 3 (3) | 0 (0)
AGE-RELATED MACULAR DEGENERATION (Eye disorders) | 0 (0) | 2 (2) | 1 (1)
OPTIC ISCHAEMIC NEUROPATHY (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
RETINAL DETACHMENT (Eye disorders) | 3 (4) | 2 (2) | 5 (7)
RETINAL VEIN OCCLUSION (Eye disorders) | 0 (0) | 2 (2) | 1 (1)
AMAUROSIS FUGAX (Eye disorders) | 0 (0) | 1 (2) | 1 (2)
ANGLE CLOSURE GLAUCOMA (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
BLINDNESS (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
CATARACT NUCLEAR (Eye disorders) | 1 (2) | 1 (1) | 0 (0)
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 1 (1) | 1 (1) | 1 (1)
CORNEAL DEGENERATION (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
ENTROPION (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
EYE HAEMORRHAGE (Eye disorders) | 3 (3) | 1 (1) | 2 (2)
MACULAR OEDEMA (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
RETINAL ARTERY EMBOLISM (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
RETINAL ARTERY OCCLUSION (Eye disorders) | 1 (2) | 1 (1) | 4 (4)
RETINAL HAEMORRHAGE (Eye disorders) | 6 (7) | 1 (1) | 2 (2)
RETINOPATHY (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
SCOTOMA (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
AMBLYOPIA (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
APHAKIA (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
ARTERIOSCLEROTIC RETINOPATHY (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
BLEPHARITIS (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
CHOROIDAL HAEMORRHAGE (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
CONJUNCTIVITIS (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
CORNEAL DECOMPENSATION (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
DIABETIC RETINOPATHY (Eye disorders) | 5 (6) | 0 (0) | 1 (2)
DIPLOPIA (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
EYELID PTOSIS (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
FUCHS' SYNDROME (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
KERATOPATHY (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
LACRIMATION INCREASED (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
LENS DISLOCATION (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
MACULAR DEGENERATION (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
MACULAR FIBROSIS (Eye disorders) | 0 (0) | 0 (0) | 2 (3)
MACULAR HOLE (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
MACULOPATHY (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
OPEN ANGLE GLAUCOMA (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
PANOPHTHALMITIS (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
PAPILLOEDEMA (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
PTERYGIUM (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
RETINAL ARTERY THROMBOSIS (Eye disorders) | 2 (3) | 0 (0) | 1 (2)
RETINAL VASCULAR THROMBOSIS (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
RETINAL VEIN THROMBOSIS (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
SCLERAL HAEMORRHAGE (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
SCLERITIS (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
STRABISMUS (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
ULCERATIVE KERATITIS (Eye disorders) | 2 (2) | 0 (0) | 1 (1)
VISUAL IMPAIRMENT (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 11 (11) | 15 (16) | 15 (17)
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 7 (9) | 5 (6) | 4 (5)
VESTIBULAR DISORDER (Ear and labyrinth disorders) | 2 (2) | 2 (2) | 0 (0)
HYPOACUSIS (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
MENIERE'S DISEASE (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
TYMPANIC MEMBRANE PERFORATION (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
DEAFNESS NEUROSENSORY (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
DEAFNESS UNILATERAL (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 1 (1)
SUDDEN HEARING LOSS (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 371 (534) | 318 (458) | 300 (418)
ATRIAL FIBRILLATION (Cardiac disorders) | 343 (495) | 315 (466) | 367 (534)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 291 (406) | 291 (421) | 270 (374)
MYOCARDIAL INFARCTION (Cardiac disorders) | 142 (154) | 147 (164) | 189 (204)
ANGINA UNSTABLE (Cardiac disorders) | 137 (154) | 127 (141) | 120 (146)
ANGINA PECTORIS (Cardiac disorders) | 80 (88) | 61 (64) | 77 (80)
SICK SINUS SYNDROME (Cardiac disorders) | 67 (68) | 50 (51) | 64 (65)
BRADYCARDIA (Cardiac disorders) | 56 (58) | 44 (47) | 40 (41)
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 38 (41) | 44 (55) | 46 (65)
ATRIAL FLUTTER (Cardiac disorders) | 46 (62) | 35 (44) | 41 (48)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 41 (44) | 33 (38) | 39 (47)
CARDIAC ARREST (Cardiac disorders) | 26 (27) | 27 (27) | 21 (23)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 28 (31) | 27 (29) | 23 (27)
CORONARY ARTERY DISEASE (Cardiac disorders) | 36 (38) | 27 (30) | 27 (27)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 22 (22) | 23 (23) | 18 (18)
ARRHYTHMIA (Cardiac disorders) | 13 (13) | 16 (17) | 13 (14)
CARDIOMYOPATHY (Cardiac disorders) | 9 (9) | 13 (13) | 7 (11)
CARDIOGENIC SHOCK (Cardiac disorders) | 15 (15) | 12 (12) | 18 (18)
BRADYARRHYTHMIA (Cardiac disorders) | 10 (10) | 11 (11) | 10 (10)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 6 (8) | 11 (11) | 12 (13)
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 6 (6) | 10 (11) | 4 (4)
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 4 (6) | 10 (12) | 4 (4)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 7 (8) | 10 (13) | 7 (10)
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 14 (14) | 9 (9) | 17 (19)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 11 (11) | 9 (11) | 7 (7)
ACUTE LEFT VENTRICULAR FAILURE (Cardiac disorders) | 4 (5) | 8 (8) | 4 (5)
CONGESTIVE CARDIOMYOPATHY (Cardiac disorders) | 10 (13) | 7 (7) | 12 (13)
CORONARY ARTERY STENOSIS (Cardiac disorders) | 5 (7) | 6 (7) | 5 (5)
PALPITATIONS (Cardiac disorders) | 6 (6) | 6 (6) | 3 (3)
SINUS BRADYCARDIA (Cardiac disorders) | 9 (9) | 6 (6) | 6 (6)
TACHYARRHYTHMIA (Cardiac disorders) | 8 (9) | 6 (6) | 15 (19)
AORTIC VALVE STENOSIS (Cardiac disorders) | 5 (6) | 5 (5) | 6 (6)
ATRIAL THROMBOSIS (Cardiac disorders) | 7 (7) | 5 (5) | 7 (7)
PERICARDIAL EFFUSION (Cardiac disorders) | 5 (5) | 5 (6) | 2 (2)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 2 (2) | 4 (5) | 2 (2)
ATRIAL TACHYCARDIA (Cardiac disorders) | 7 (8) | 4 (5) | 6 (9)
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 12 (12) | 4 (4) | 22 (23)
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 0 (0) | 4 (4) | 3 (3)
CARDIOPULMONARY FAILURE (Cardiac disorders) | 4 (4) | 4 (4) | 8 (9)
CORONARY ARTERY INSUFFICIENCY (Cardiac disorders) | 1 (1) | 4 (4) | 1 (1)
ISCHAEMIC CARDIOMYOPATHY (Cardiac disorders) | 7 (8) | 4 (4) | 4 (4)
MYOCARDIAL FIBROSIS (Cardiac disorders) | 3 (3) | 4 (4) | 1 (1)
RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 7 (9) | 4 (4) | 2 (2)
ADAMS-STOKES SYNDROME (Cardiac disorders) | 0 (0) | 3 (3) | 2 (2)
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 6 (6) | 3 (3) | 3 (3)
PERICARDIAL HAEMORRHAGE (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0)
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 7 (7) | 3 (3) | 3 (3)
AORTIC VALVE DISEASE (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
AORTIC VALVE INCOMPETENCE (Cardiac disorders) | 2 (2) | 2 (2) | 2 (2)
CARDIAC VALVE DISEASE (Cardiac disorders) | 5 (5) | 2 (2) | 3 (4)
CARDIOVASCULAR INSUFFICIENCY (Cardiac disorders) | 3 (3) | 2 (2) | 4 (4)
COR PULMONALE (Cardiac disorders) | 2 (2) | 2 (2) | 1 (2)
HEART VALVE INCOMPETENCE (Cardiac disorders) | 4 (5) | 2 (2) | 2 (2)
HYPERTROPHIC CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
STRESS CARDIOMYOPATHY (Cardiac disorders) | 2 (2) | 2 (2) | 1 (1)
SUPRAVENTRICULAR TACHYARRHYTHMIA (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 2 (2) | 2 (2) | 5 (5)
TRICUSPID VALVE INCOMPETENCE (Cardiac disorders) | 2 (2) | 2 (2) | 2 (2)
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 3 (3) | 2 (2) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
AORTIC VALVE CALCIFICATION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
BIFASCICULAR BLOCK (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
BUNDLE BRANCH BLOCK LEFT (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
CARDIAC ASTHMA (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
CARDIAC DISORDER (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
CARDIORENAL SYNDROME (Cardiac disorders) | 0 (0) | 1 (2) | 1 (1)
CARDIOVASCULAR DISORDER (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
CHORDAE TENDINAE RUPTURE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CHRONOTROPIC INCOMPETENCE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CONDUCTION DISORDER (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
CORONARY ARTERY ANEURYSM (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
DRESSLER'S SYNDROME (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERTENSIVE HEART DISEASE (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
INTRACARDIAC THROMBUS (Cardiac disorders) | 6 (6) | 1 (1) | 0 (0)
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 5 (5) | 1 (1) | 3 (3)
MITRAL VALVE DISEASE (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
MITRAL VALVE STENOSIS (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
PULSELESS ELECTRICAL ACTIVITY (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
RHEUMATIC HEART DISEASE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
SUPRAVENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
VENTRICULAR TACHYARRHYTHMIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
AORTIC VALVE DISEASE MIXED (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
ARRHYTHMIA SUPRAVENTRICULAR (Cardiac disorders) | 2 (2) | 0 (0) | 2 (2)
BUNDLE BRANCH BLOCK RIGHT (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
CARDIAC FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
CARDIAC TAMPONADE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
COR PULMONALE ACUTE (Cardiac disorders) | 0 (0) | 0 (0) | 2 (4)
CORONARY ARTERY EMBOLISM (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
CORONARY ARTERY THROMBOSIS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
CYTOTOXIC CARDIOMYOPATHY (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
DIASTOLIC DYSFUNCTION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
ENDOCARDITIS NONINFECTIVE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
METABOLIC CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
MITRAL VALVE PROLAPSE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
NODAL ARRHYTHMIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
PERICARDITIS (Cardiac disorders) | 4 (4) | 0 (0) | 4 (4)
PRINZMETAL ANGINA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
RHYTHM IDIOVENTRICULAR (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
SINUS ARREST (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
SINUS ARRHYTHMIA (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
SYSTOLIC DYSFUNCTION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
TACHYCARDIA PAROXYSMAL (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
TORSADE DE POINTES (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
TRIFASCICULAR BLOCK (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
WOLFF-PARKINSON-WHITE SYNDROME (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 29 (32) | 42 (46) | 36 (38)
HYPOTENSION (Vascular disorders) | 23 (23) | 24 (25) | 30 (30)
DEEP VEIN THROMBOSIS (Vascular disorders) | 20 (21) | 17 (18) | 11 (13)
HYPERTENSIVE CRISIS (Vascular disorders) | 15 (15) | 16 (16) | 13 (14)
AORTIC ANEURYSM (Vascular disorders) | 12 (12) | 9 (9) | 14 (15)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 11 (12) | 9 (9) | 24 (28)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 5 (6) | 9 (10) | 13 (15)
AORTIC STENOSIS (Vascular disorders) | 15 (15) | 8 (8) | 10 (10)
ARTERIOSCLEROSIS (Vascular disorders) | 7 (7) | 8 (8) | 4 (4)
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 6 (6) | 8 (12) | 5 (7)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 9 (11) | 7 (8) | 9 (9)
ARTERIOSCLEROSIS OBLITERANS (Vascular disorders) | 1 (1) | 5 (6) | 1 (1)
AORTIC ANEURYSM RUPTURE (Vascular disorders) | 5 (5) | 4 (4) | 4 (4)
BLEEDING VARICOSE VEIN (Vascular disorders) | 0 (0) | 4 (4) | 0 (0)
VARICOSE VEIN (Vascular disorders) | 1 (1) | 4 (4) | 4 (4)
AORTIC DISSECTION (Vascular disorders) | 2 (2) | 3 (3) | 2 (2)
FEMORAL ARTERIAL STENOSIS (Vascular disorders) | 3 (3) | 3 (3) | 2 (2)
HAEMORRHAGE (Vascular disorders) | 2 (2) | 3 (4) | 0 (0)
HYPERTENSIVE EMERGENCY (Vascular disorders) | 1 (1) | 3 (3) | 2 (2)
PERIPHERAL EMBOLISM (Vascular disorders) | 3 (4) | 3 (3) | 7 (8)
THROMBOSIS (Vascular disorders) | 1 (1) | 3 (3) | 2 (2)
ARTERIAL DISORDER (Vascular disorders) | 0 (0) | 2 (3) | 2 (2)
ARTERIAL THROMBOSIS LIMB (Vascular disorders) | 6 (6) | 2 (2) | 3 (4)
ARTERITIS OBLITERANS (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
DISTRIBUTIVE SHOCK (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
EXTREMITY NECROSIS (Vascular disorders) | 5 (5) | 2 (2) | 4 (4)
FEMORAL ARTERY EMBOLISM (Vascular disorders) | 3 (3) | 2 (3) | 1 (1)
INTRA-ABDOMINAL HAEMATOMA (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
SUBCLAVIAN VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
VENOUS INSUFFICIENCY (Vascular disorders) | 0 (0) | 2 (2) | 4 (4)
VENOUS THROMBOSIS (Vascular disorders) | 2 (2) | 2 (2) | 1 (1)
VENOUS THROMBOSIS LIMB (Vascular disorders) | 1 (1) | 2 (2) | 2 (2)
AORTIC DILATATION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
AORTIC THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 2 (2) | 1 (1) | 6 (6)
ARTERIAL THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1) | 2 (2)
CIRCULATORY COLLAPSE (Vascular disorders) | 3 (3) | 1 (1) | 3 (3)
DIABETIC MACROANGIOPATHY (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
DIABETIC VASCULAR DISORDER (Vascular disorders) | 0 (0) | 1 (3) | 0 (0)
EMBOLISM ARTERIAL (Vascular disorders) | 6 (7) | 1 (1) | 1 (2)
EXTRAVASATION BLOOD (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
FEMORAL ARTERY ANEURYSM (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
HAEMATOMA (Vascular disorders) | 4 (4) | 1 (1) | 0 (0)
HYPOVOLAEMIC SHOCK (Vascular disorders) | 5 (5) | 1 (1) | 1 (1)
ILIAC ARTERY EMBOLISM (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
INFARCTION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
INTERMITTENT CLAUDICATION (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
ISCHAEMIA (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
LYMPHATIC FISTULA (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
LYMPHOCELE (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
LYMPHOEDEMA (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
PERIPHERAL ARTERY ANEURYSM (Vascular disorders) | 1 (1) | 1 (1) | 3 (3)
RHEUMATOID VASCULITIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
SHOCK HAEMORRHAGIC (Vascular disorders) | 1 (1) | 1 (1) | 3 (3)
SUBCLAVIAN STEAL SYNDROME (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
SUPERIOR MESENTERIC ARTERY SYNDROME (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
THROMBOPHLEBITIS (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
VARICOSE ULCERATION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
VASCULAR INSUFFICIENCY (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
VASCULITIS (Vascular disorders) | 0 (0) | 1 (2) | 3 (3)
ACCELERATED HYPERTENSION (Vascular disorders) | 6 (6) | 0 (0) | 4 (6)
ANEURYSM (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
ANEURYSM RUPTURED (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
ANGIOPATHY (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
AORTIC DISSECTION RUPTURE (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
AORTIC EMBOLUS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
AORTIC RUPTURE (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
ARTERIAL HAEMORRHAGE (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
ARTERIAL STENOSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
ARTERIAL STENOSIS LIMB (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
ARTERIOSCLEROSIS MOENCKEBERG-TYPE (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
EMBOLISM (Vascular disorders) | 1 (1) | 0 (0) | 3 (3)
ESSENTIAL HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
FIBROMUSCULAR DYSPLASIA (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
HAEMODYNAMIC INSTABILITY (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
ILIAC ARTERY STENOSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
ILIAC ARTERY THROMBOSIS (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
LABILE HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
POOR PERIPHERAL CIRCULATION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
SHOCK (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
TEMPORAL ARTERITIS (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
THROMBOANGIITIS OBLITERANS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
THROMBOPHLEBITIS SUPERFICIAL (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
THROMBOSED VARICOSE VEIN (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
VENOUS HAEMORRHAGE (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 89 (127) | 93 (125) | 105 (150)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 48 (56) | 36 (42) | 18 (18)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 20 (21) | 29 (29) | 26 (26)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 18 (19) | 26 (27) | 20 (24)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 26 (28) | 21 (22) | 26 (26)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 19 (19) | 20 (23) | 17 (17)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 20 (23) | 10 (10)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 19 (22) | 14 (16) | 23 (24)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 19 (28) | 13 (13) | 19 (22)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 14 (15) | 13 (13) | 21 (24)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 12 (14) | 12 (12)
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 11 (12) | 8 (8)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 9 (11) | 8 (8)
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (7) | 6 (7)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6) | 7 (9)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 6 (6) | 5 (6)
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5) | 4 (4)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 4 (4)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) | 3 (3)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 1 (1)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 3 (4)
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 2 (2)
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4) | 2 (2)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
BRONCHIECTASIS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 1 (1)
CHRONIC RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 4 (4)
ORGANISING PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2)
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1)
PULMONARY TOXICITY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
ASPHYXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
BRONCHIAL HYPERREACTIVITY (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
BRONCHOPNEUMOPATHY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
DYSPNOEA AT REST (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 8 (9)
EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
FOREIGN BODY ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOVENTILATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
NASAL POLYPS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
PULMONARY INFARCTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
THORACIC HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
VOCAL CORD CYST (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
VOCAL CORD INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
ALLERGIC GRANULOMATOUS ANGIITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
ALVEOLITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
ASTHMATIC CRISIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
BRONCHIAL HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
BRONCHIAL SECRETION RETENTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
BRONCHITIS CHRONIC (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
BRONCHOMALACIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
CHOKING (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
DIAPHRAGMATIC HERNIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
HYDROPNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
HYDROTHORAX (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1)
HYPERCAPNIA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
LARYNGEAL DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
LARYNGEAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
NASAL CYST (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
NASAL SEPTUM DEVIATION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
NOCTURNAL DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OBSTRUCTIVE AIRWAYS DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PHARYNGEAL HAEMATOMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PHARYNGEAL HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PHARYNGEAL MASS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PICKWICKIAN SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 0 (0)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
PULMONARY ALVEOLAR HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PULMONARY ARTERIAL HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2)
PULMONARY ARTERY THROMBOSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
PULMONARY GRANULOMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
RESPIRATORY ACIDOSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
RESPIRATORY TRACT HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
SINUS POLYP (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
TRACHEAL MASS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
VOCAL CORD POLYP (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 83 (85) | 89 (97) | 59 (64)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 24 (28) | 42 (44) | 28 (30)
INGUINAL HERNIA (Gastrointestinal disorders) | 24 (25) | 33 (37) | 36 (36)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 28 (32) | 29 (33) | 38 (41)
GASTRITIS (Gastrointestinal disorders) | 11 (12) | 27 (28) | 12 (12)
MELAENA (Gastrointestinal disorders) | 8 (9) | 26 (27) | 7 (8)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 22 (23) | 19 (19) | 13 (13)
COLONIC POLYP (Gastrointestinal disorders) | 9 (10) | 18 (19) | 16 (17)
DIARRHOEA (Gastrointestinal disorders) | 17 (17) | 17 (17) | 7 (7)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 13 (14) | 14 (14) | 19 (27)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 9 (13) | 14 (16) | 11 (12)
HAEMATOCHEZIA (Gastrointestinal disorders) | 8 (8) | 13 (13) | 10 (10)
PANCREATITIS (Gastrointestinal disorders) | 23 (23) | 13 (14) | 6 (6)
ILEUS (Gastrointestinal disorders) | 6 (6) | 11 (12) | 6 (7)
GASTRITIS EROSIVE (Gastrointestinal disorders) | 2 (2) | 10 (10) | 10 (10)
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 6 (6) | 10 (11) | 3 (3)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 8 (8) | 10 (11) | 4 (4)
ABDOMINAL PAIN (Gastrointestinal disorders) | 9 (10) | 9 (10) | 11 (12)
CONSTIPATION (Gastrointestinal disorders) | 13 (14) | 9 (9) | 5 (5)
DYSPEPSIA (Gastrointestinal disorders) | 4 (4) | 8 (8) | 4 (4)
UMBILICAL HERNIA (Gastrointestinal disorders) | 6 (6) | 8 (8) | 2 (2)
HAEMATEMESIS (Gastrointestinal disorders) | 7 (7) | 7 (7) | 2 (2)
HAEMORRHOIDS (Gastrointestinal disorders) | 3 (3) | 7 (7) | 6 (6)
DUODENAL ULCER (Gastrointestinal disorders) | 3 (3) | 6 (7) | 3 (3)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 6 (6) | 6 (6) | 5 (5)
GASTRIC ULCER (Gastrointestinal disorders) | 13 (14) | 5 (6) | 11 (11)
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 9 (9) | 5 (5) | 8 (8)
GASTRITIS HAEMORRHAGIC (Gastrointestinal disorders) | 1 (1) | 5 (5) | 0 (0)
VOMITING (Gastrointestinal disorders) | 3 (3) | 5 (6) | 4 (4)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 4 (4) | 4 (4) | 6 (7)
ABDOMINAL STRANGULATED HERNIA (Gastrointestinal disorders) | 0 (0) | 4 (4) | 2 (2)
ASCITES (Gastrointestinal disorders) | 3 (3) | 4 (4) | 3 (3)
COLITIS (Gastrointestinal disorders) | 5 (6) | 4 (4) | 6 (6)
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 5 (5) | 4 (4) | 1 (1)
GASTRIC POLYPS (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1)
INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 4 (4) | 4 (5) | 0 (0)
LARGE INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 4 (4) | 4 (4) | 2 (2)
ABDOMINAL HERNIA (Gastrointestinal disorders) | 3 (3) | 3 (3) | 3 (3)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 4 (4) | 3 (3) | 2 (2)
DENTAL CARIES (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
DIVERTICULUM (Gastrointestinal disorders) | 3 (3) | 3 (3) | 1 (1)
FAECALOMA (Gastrointestinal disorders) | 2 (2) | 3 (4) | 3 (3)
FAECES DISCOLOURED (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0)
GASTRIC ANTRAL VASCULAR ECTASIA (Gastrointestinal disorders) | 1 (1) | 3 (4) | 0 (0)
HIATUS HERNIA (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (4)
INGUINAL HERNIA STRANGULATED (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (2)
PANCREATIC MASS (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
PERIODONTITIS (Gastrointestinal disorders) | 3 (3) | 3 (3) | 7 (7)
RETROPERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 5 (5) | 3 (3) | 2 (2)
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2)
CAECITIS (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
DIARRHOEA HAEMORRHAGIC (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (4)
DIVERTICULUM INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 7 (7) | 2 (2) | 2 (2)
DYSPHAGIA (Gastrointestinal disorders) | 5 (6) | 2 (2) | 2 (2)
FEMORAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
GASTROINTESTINAL VASCULAR MALFORMATION (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
INGUINAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 4 (4) | 2 (2) | 5 (5)
INTESTINAL POLYP (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
PEPTIC ULCER (Gastrointestinal disorders) | 6 (6) | 2 (2) | 1 (1)
PEPTIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
POLYP COLORECTAL (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
UMBILICAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2)
ABDOMINAL ADHESIONS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2)
ABDOMINAL HERNIA OBSTRUCTIVE (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
ANAL FISSURE (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
CHRONIC GASTROINTESTINAL BLEEDING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
COLITIS MICROSCOPIC (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
COLONIC STENOSIS (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
CROHN'S DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
DIVERTICULUM INTESTINAL (Gastrointestinal disorders) | 3 (3) | 1 (1) | 5 (5)
DUODENAL POLYP (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
DUODENITIS (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
ENTEROCOLITIS HAEMORRHAGIC (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
FAECAL INCONTINENCE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
FEMORAL HERNIA (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
GASTRIC DYSPLASIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
GASTRIC MUCOSAL LESION (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
GASTRITIS ATROPHIC (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
GASTRODUODENITIS (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
GASTROINTESTINAL INFLAMMATION (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
GASTROINTESTINAL TOXICITY (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0)
GASTROINTESTINAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
GLOSSITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
HAEMORRHAGIC EROSIVE GASTRITIS (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
ILEUS PARALYTIC (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (3)
INFLAMMATORY BOWEL DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 2 (2) | 1 (1) | 6 (6)
INTESTINAL MASS (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
INTESTINAL POLYP HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
INTESTINAL STENOSIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (3)
OESOPHAGEAL FOOD IMPACTION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OESOPHAGEAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OESOPHAGEAL RUPTURE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OESOPHAGEAL SPASM (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
OESOPHAGEAL STENOSIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
OESOPHAGEAL ULCER (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (1)
OESOPHAGITIS (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0)
PANCREATIC NECROSIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
PANCREATITIS CHRONIC (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
PANCREATITIS NECROTISING (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1)
PERIODONTAL DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
PNEUMOPERITONEUM (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
PROTEIN-LOSING GASTROENTEROPATHY (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
PYLORUS DILATATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
RADICULAR CYST (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
RECTAL POLYP (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
RECTAL ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
REFLUX GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
RETROPERITONEAL HAEMATOMA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL MASS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL WALL HAEMATOMA (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0)
ACUTE ABDOMEN (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
ALCOHOLIC PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
ANAL FISTULA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
ANAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
COELIAC DISEASE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
COLON DYSPLASIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
COLONIC FISTULA (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
COLONIC PSEUDO-OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
DIABETIC GASTROPATHY (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
DIVERTICULITIS INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
DIVERTICULUM OESOPHAGEAL (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
ENTERITIS (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
ENTEROCOLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
ENTEROVESICAL FISTULA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
FOOD POISONING (Gastrointestinal disorders) | 4 (4) | 0 (0) | 2 (2)
GASTRIC VARICES (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GASTRODUODENAL ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GASTROINTESTINAL DYSPLASIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GASTROINTESTINAL HYPOMOTILITY (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GASTROINTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GASTROINTESTINAL NECROSIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
GASTROINTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GASTROINTESTINAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GASTROPLEURAL FISTULA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GIANT CELL EPULIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ILEITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
INTESTINAL HAEMATOMA (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
INTESTINAL INFARCTION (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
LARGE INTESTINAL ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
LIP HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
MALLORY-WEISS SYNDROME (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
MESENTERIC ARTERY EMBOLISM (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
MESENTERIC ARTERY THROMBOSIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
MESENTERIC VEIN THROMBOSIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
MOUTH ULCERATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
ODYNOPHAGIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OESOPHAGEAL ACHALASIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
ORAL DYSAESTHESIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
PANCREATIC CYST (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
PANCREATITIS RELAPSING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
PANCREATOLITHIASIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
PAROTID GLAND INFLAMMATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
PERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
PNEUMATOSIS INTESTINALIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
POOR DENTAL CONDITION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
PROCTALGIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
RECTAL PROLAPSE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
SALIVARY GLAND CALCULUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
SMALL INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3)
SMALL INTESTINAL PERFORATION (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
SPIGELIAN HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
SUBILEUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
TONGUE CYST (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
TOOTHACHE (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
VARICES OESOPHAGEAL (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
VOLVULUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 25 (27) | 26 (27) | 31 (31)
CHOLECYSTITIS (Hepatobiliary disorders) | 23 (23) | 25 (27) | 15 (15)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 18 (18) | 22 (23) | 18 (20)
BILE DUCT STONE (Hepatobiliary disorders) | 15 (15) | 9 (10) | 11 (12)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 4 (4) | 7 (7) | 9 (9)
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 3 (3) | 5 (5) | 2 (2)
JAUNDICE (Hepatobiliary disorders) | 0 (0) | 4 (4) | 3 (3)
AUTOIMMUNE HEPATITIS (Hepatobiliary disorders) | 0 (0) | 3 (3) | 0 (0)
HEPATITIS CHRONIC ACTIVE (Hepatobiliary disorders) | 0 (0) | 3 (4) | 0 (0)
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 0 (0) | 2 (3) | 0 (0)
BILIARY COLIC (Hepatobiliary disorders) | 2 (2) | 2 (2) | 2 (2)
CHOLANGITIS (Hepatobiliary disorders) | 2 (2) | 2 (2) | 4 (4)
HEPATIC FAILURE (Hepatobiliary disorders) | 4 (4) | 2 (3) | 1 (1)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 3 (3) | 2 (2) | 2 (2)
ISCHAEMIC HEPATITIS (Hepatobiliary disorders) | 1 (1) | 2 (2) | 2 (2)
ACUTE HEPATIC FAILURE (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0)
ALCOHOLIC LIVER DISEASE (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
BILIARY FISTULA (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
CHOLANGITIS ACUTE (Hepatobiliary disorders) | 2 (2) | 1 (1) | 2 (2)
GALLBLADDER POLYP (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
HEPATIC CYST (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1)
HEPATIC CYST RUPTURED (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
HEPATIC STEATOSIS (Hepatobiliary disorders) | 3 (3) | 1 (1) | 3 (3)
HEPATITIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 4 (4)
HEPATOTOXICITY (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
HYDROCHOLECYSTIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
JAUNDICE CHOLESTATIC (Hepatobiliary disorders) | 6 (6) | 1 (1) | 5 (5)
AMPULLA OF VATER STENOSIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
BILE DUCT STENOSIS (Hepatobiliary disorders) | 2 (3) | 0 (0) | 0 (0)
BILIARY DYSKINESIA (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
CHOLELITHIASIS OBSTRUCTIVE (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0)
CHOLESTASIS (Hepatobiliary disorders) | 4 (4) | 0 (0) | 1 (1)
CHRONIC HEPATIC FAILURE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
GALLBLADDER DISORDER (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
HAEMOBILIA (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
HEPATIC CONGESTION (Hepatobiliary disorders) | 2 (2) | 0 (0) | 2 (3)
HEPATIC ISCHAEMIA (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
HEPATITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 0 (0) | 2 (2)
HEPATITIS ALCOHOLIC (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
HEPATITIS TOXIC (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
HEPATOMEGALY (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
HEPATORENAL FAILURE (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
HEPATORENAL SYNDROME (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
LIVER DISORDER (Hepatobiliary disorders) | 1 (1) | 0 (0) | 2 (2)
LIVER INJURY (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
PORTAL VEIN THROMBOSIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
POST CHOLECYSTECTOMY SYNDROME (Hepatobiliary disorders) | 2 (2) | 0 (0) | 1 (1)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 12 (13) | 6 (6) | 14 (14)
SKIN HAEMORRHAGE (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5) | 4 (4)
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 1 (1)
DERMAL CYST (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
DERMATOMYOSITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 2 (2)
DRUG RASH WITH EOSINOPHILIA AND SYSTEMIC SYMPTOMS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
DRY GANGRENE (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERKERATOSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
PURPURA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
SKIN NECROSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
STASIS DERMATITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
STEVENS-JOHNSON SYNDROME (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
ACANTHOSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
CUTANEOUS LUPUS ERYTHEMATOSUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
DERMATITIS (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
ECZEMA (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0)
ECZEMA NUMMULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
GRANULOMA SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
HAEMORRHAGE SUBCUTANEOUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
HENOCH-SCHONLEIN PURPURA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
LEUKOCYTOCLASTIC VASCULITIS (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
NEURODERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
PANNICULITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
PEMPHIGOID (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
PRURIGO (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
SCAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
SEBORRHOEIC DERMATITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
SKIN ULCER HAEMORRHAGE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
SUBCUTANEOUS NODULE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
SWELLING FACE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 62 (69) | 70 (78) | 61 (65)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 14 (14) | 16 (17) | 12 (12)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 6 (6) | 13 (13) | 10 (11)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 11 (12) | 8 (11) | 9 (10)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 6 (6) | 7 (9) | 8 (8)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (7) | 7 (7)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 15 (16) | 5 (5) | 7 (9)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5) | 3 (3)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 10 (13) | 5 (5) | 4 (4)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5) | 1 (1)
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5) | 14 (15)
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 0 (0)
HAEMARTHROSIS (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3) | 1 (1)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1)
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 9 (10) | 3 (3) | 14 (16)
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0)
GOUTY ARTHRITIS (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 7 (9)
INTERVERTEBRAL DISC DISORDER (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (3) | 0 (0)
POLYARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 2 (2)
ANKYLOSING SPONDYLITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
AXILLARY MASS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
BURSITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2)
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
CHONDROCALCINOSIS PYROPHOSPHATE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
INCLUSION BODY MYOSITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
JOINT INSTABILITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (3) | 3 (3)
MYOSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OSTEOPOROTIC FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
PERIARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
PERIOSTITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
POLYMYALGIA RHEUMATICA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 5 (5)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 7 (7)
SPONDYLITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
SPONDYLOARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (3)
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
TORTICOLLIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
TRIGGER FINGER (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (2)
ARTICULAR CALCIFICATION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
BACK DISORDER (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
BONE CYST (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
CHONDROPATHY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
DEFORMITY THORAX (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
DUPUYTREN'S CONTRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (4)
EXOSTOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
FASCIITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
FISTULA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 5 (5)
FRACTURE MALUNION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
GOUTY TOPHUS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC COMPRESSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (4)
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
LATERAL PATELLAR COMPRESSION SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
MUSCLE ATROPHY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
MUSCLE DISORDER (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
MUSCLE HAEMORRHAGE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 5 (5)
MUSCLE TWITCHING (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
MYOPATHY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
NEUROPATHIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
OSTEITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OSTEOCHONDROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 4 (5)
OSTEONECROSIS OF JAW (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
SCOLIOSIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
SPINAL DISORDER (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
SYMPATHETIC POSTERIOR CERVICAL SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
UNDIFFERENTIATED CONNECTIVE TISSUE DISEASE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 64 (67) | 68 (71) | 57 (60)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 63 (68) | 53 (56) | 62 (67)
RENAL FAILURE (Renal and urinary disorders) | 29 (30) | 29 (30) | 16 (17)
NEPHROLITHIASIS (Renal and urinary disorders) | 7 (8) | 17 (19) | 7 (8)
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 14 (15) | 13 (14) | 12 (14)
CALCULUS URETERIC (Renal and urinary disorders) | 2 (2) | 9 (9) | 8 (8)
URINARY RETENTION (Renal and urinary disorders) | 3 (3) | 7 (7) | 9 (9)
CALCULUS URINARY (Renal and urinary disorders) | 4 (4) | 6 (7) | 2 (2)
RENAL IMPAIRMENT (Renal and urinary disorders) | 7 (8) | 6 (6) | 13 (15)
ACUTE PRERENAL FAILURE (Renal and urinary disorders) | 5 (5) | 5 (5) | 0 (0)
RENAL CYST (Renal and urinary disorders) | 1 (1) | 4 (5) | 2 (2)
URETHRAL STENOSIS (Renal and urinary disorders) | 4 (4) | 4 (4) | 2 (2)
CALCULUS BLADDER (Renal and urinary disorders) | 3 (3) | 3 (3) | 1 (1)
DIABETIC NEPHROPATHY (Renal and urinary disorders) | 1 (1) | 3 (3) | 1 (1)
RENAL ARTERY STENOSIS (Renal and urinary disorders) | 0 (0) | 3 (3) | 2 (2)
STAG HORN CALCULUS (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0)
RENAL COLIC (Renal and urinary disorders) | 2 (2) | 2 (2) | 3 (3)
RENAL INFARCT (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
URINARY INCONTINENCE (Renal and urinary disorders) | 3 (3) | 2 (2) | 1 (2)
AZOTAEMIA (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2)
BLADDER MASS (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
BLADDER STENOSIS (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
BLADDER TAMPONADE (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
CYSTITIS GLANDULARIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
CYSTITIS HAEMORRHAGIC (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
DYSURIA (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
HYDRONEPHROSIS (Renal and urinary disorders) | 2 (2) | 1 (1) | 5 (5)
NEPHROPATHY (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2)
NEPHROSCLEROSIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
NEPHROTIC SYNDROME (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
OBSTRUCTIVE UROPATHY (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
POLLAKIURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
POLYURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
RENAL INJURY (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
STRESS URINARY INCONTINENCE (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
TUBULOINTERSTITIAL NEPHRITIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
URETHRAL HAEMORRHAGE (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
URINARY BLADDER POLYP (Renal and urinary disorders) | 1 (2) | 1 (2) | 1 (1)
URINARY TRACT DISORDER (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
BLADDER OUTLET OBSTRUCTION (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2)
BLADDER PROLAPSE (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
CYSTITIS NONINFECTIVE (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
GLOMERULONEPHRITIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
GLOMERULONEPHROPATHY (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
HAEMORRHAGE URINARY TRACT (Renal and urinary disorders) | 2 (2) | 0 (0) | 2 (2)
HYPERTENSIVE NEPHROPATHY (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
NEPHRITIS AUTOIMMUNE (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
NEUROGENIC BLADDER (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
RENAL MASS (Renal and urinary disorders) | 1 (1) | 0 (0) | 3 (3)
RENAL TUBULAR NECROSIS (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
URETERIC STENOSIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
URETHRAL DISCHARGE (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
URETHRAL OBSTRUCTION (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
URETHRAL POLYP (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
URINARY BLADDER HAEMORRHAGE (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
UROGENITAL HAEMORRHAGE (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 35 (37) | 29 (31) | 17 (18)
PROSTATITIS (Reproductive system and breast disorders) | 6 (7) | 5 (5) | 2 (2)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 7 (7) | 4 (4) | 3 (3)
METRORRHAGIA (Reproductive system and breast disorders) | 3 (3) | 3 (3) | 1 (1)
PROSTATOMEGALY (Reproductive system and breast disorders) | 1 (1) | 3 (3) | 2 (2)
UTERINE POLYP (Reproductive system and breast disorders) | 1 (1) | 3 (3) | 1 (1)
BREAST MASS (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
CERVIX HAEMORRHAGE UTERINE (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
ACQUIRED HYDROCELE (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 2 (2)
ACQUIRED PHIMOSIS (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 2 (2)
BALANITIS (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
CERVICAL POLYP (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
CERVIX HAEMATOMA UTERINE (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
COLPOCELE (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
ENDOMETRIAL HYPERPLASIA (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
EPIDIDYMITIS (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0)
GENITAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
OVARIAN CYST (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 2 (2)
POSTMENOPAUSAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
PROSTATISM (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
RECTOCELE (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 7 (7)
UTERINE PROLAPSE (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 1 (1)
BREAST CALCIFICATIONS (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
BREAST CYST (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2)
BREAST PAIN (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
ENDOMETRIAL HYPERTROPHY (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 1 (1)
ENDOMETRIOSIS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
FEMALE GENITAL TRACT FISTULA (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
GYNAECOMASTIA (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
OVARIAN MASS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
PELVIC PAIN (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
PENILE HAEMORRHAGE (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
PROSTATIC DYSPLASIA (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
PROSTATIC OBSTRUCTION (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2)
SCROTAL OEDEMA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
UTERINE CYST (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
VAGINAL PROLAPSE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2)
ARTERIOVENOUS MALFORMATION (Congenital, familial and genetic disorders) | 0 (0) | 1 (2) | 0 (0)
DIVERTICULITIS MECKEL'S (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL ANGIODYSPLASIA (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL ANGIODYSPLASIA HAEMORRHAGIC (Congenital, familial and genetic disorders) | 0 (0) | 1 (2) | 0 (0)
GITELMAN'S SYNDROME (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
HAEMORRHAGIC ARTERIOVENOUS MALFORMATION (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
HIP DYSPLASIA (Congenital, familial and genetic disorders) | 1 (1) | 1 (1) | 0 (0)
HYDROCELE (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 2 (2)
ATRIAL SEPTAL DEFECT (Congenital, familial and genetic disorders) | 3 (3) | 0 (0) | 0 (0)
FRIEDREICH'S ATAXIA (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
PENOSCROTAL FUSION (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
PHIMOSIS (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
RILEY-DAY SYNDROME (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
VENTRICULAR SEPTAL DEFECT (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
DEATH (General disorders) | 91 (91) | 80 (80) | 78 (78)
NON-CARDIAC CHEST PAIN (General disorders) | 39 (40) | 50 (54) | 54 (58)
SUDDEN DEATH (General disorders) | 45 (46) | 29 (29) | 35 (35)
CHEST PAIN (General disorders) | 24 (26) | 26 (27) | 33 (35)
SUDDEN CARDIAC DEATH (General disorders) | 24 (24) | 23 (23) | 24 (24)
DEVICE DISLOCATION (General disorders) | 12 (14) | 11 (13) | 6 (7)
ASTHENIA (General disorders) | 12 (12) | 8 (8) | 17 (19)
PYREXIA (General disorders) | 6 (6) | 8 (8) | 10 (11)
CHEST DISCOMFORT (General disorders) | 7 (7) | 7 (7) | 7 (7)
MULTI-ORGAN FAILURE (General disorders) | 14 (14) | 7 (7) | 18 (18)
DEVICE BATTERY ISSUE (General disorders) | 6 (6) | 5 (5) | 8 (8)
DEVICE MALFUNCTION (General disorders) | 6 (6) | 5 (6) | 7 (7)
OEDEMA PERIPHERAL (General disorders) | 5 (5) | 5 (5) | 3 (3)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 7 (7) | 4 (4) | 7 (9)
DEVICE FAILURE (General disorders) | 4 (4) | 3 (3) | 1 (1)
FATIGUE (General disorders) | 2 (2) | 3 (3) | 1 (1)
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 2 (2) | 3 (3) | 0 (0)
ADVERSE DRUG REACTION (General disorders) | 2 (2) | 2 (2) | 0 (0)
CARDIAC DEATH (General disorders) | 5 (5) | 2 (2) | 5 (5)
GAIT DISTURBANCE (General disorders) | 2 (2) | 2 (2) | 3 (3)
MEDICAL DEVICE COMPLICATION (General disorders) | 0 (0) | 2 (2) | 2 (2)
APPLICATION SITE BLEEDING (General disorders) | 0 (0) | 1 (1) | 0 (0)
CALCINOSIS (General disorders) | 0 (0) | 1 (1) | 0 (0)
DEVICE CONNECTION ISSUE (General disorders) | 0 (0) | 1 (1) | 0 (0)
DEVICE LEAD DAMAGE (General disorders) | 0 (0) | 1 (1) | 2 (2)
DEVICE PACING ISSUE (General disorders) | 0 (0) | 1 (1) | 0 (0)
DISCOMFORT (General disorders) | 1 (1) | 1 (1) | 0 (0)
DRUG WITHDRAWAL SYNDROME (General disorders) | 0 (0) | 1 (1) | 0 (0)
GRAVITATIONAL OEDEMA (General disorders) | 0 (0) | 1 (1) | 0 (0)
HERNIA (General disorders) | 0 (0) | 1 (1) | 0 (0)
HERNIA OBSTRUCTIVE (General disorders) | 0 (0) | 1 (1) | 2 (2)
IMPAIRED HEALING (General disorders) | 0 (0) | 1 (1) | 2 (2)
IMPLANT SITE HAEMATOMA (General disorders) | 0 (0) | 1 (1) | 1 (1)
IMPLANT SITE REACTION (General disorders) | 0 (0) | 1 (1) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 1 (2) | 0 (0)
INJECTION SITE HAEMATOMA (General disorders) | 2 (2) | 1 (1) | 1 (1)
ISCHAEMIC ULCER (General disorders) | 0 (0) | 1 (1) | 1 (1)
MUCOSAL HAEMORRHAGE (General disorders) | 0 (0) | 1 (1) | 0 (0)
OEDEMA (General disorders) | 0 (0) | 1 (1) | 0 (0)
PACEMAKER SYNDROME (General disorders) | 0 (0) | 1 (1) | 0 (0)
PUNCTURE SITE HAEMORRHAGE (General disorders) | 0 (0) | 1 (1) | 0 (0)
VESSEL PUNCTURE SITE HAEMATOMA (General disorders) | 1 (1) | 1 (1) | 2 (2)
ACCIDENTAL DEATH (General disorders) | 1 (1) | 0 (0) | 0 (0)
CATHETER SITE HAEMORRHAGE (General disorders) | 1 (1) | 0 (0) | 0 (0)
DEVICE BREAKAGE (General disorders) | 2 (2) | 0 (0) | 0 (0)
DEVICE CAPTURING ISSUE (General disorders) | 1 (1) | 0 (0) | 0 (0)
DEVICE ISSUE (General disorders) | 1 (1) | 0 (0) | 0 (0)
DEVICE LEAD ISSUE (General disorders) | 3 (3) | 0 (0) | 0 (0)
DEVICE LEAKAGE (General disorders) | 0 (0) | 0 (0) | 1 (1)
DEVICE OCCLUSION (General disorders) | 0 (0) | 0 (0) | 2 (2)
DROWNING (General disorders) | 0 (0) | 0 (0) | 2 (2)
GENERALISED OEDEMA (General disorders) | 2 (2) | 0 (0) | 3 (3)
IMPLANT SITE EROSION (General disorders) | 1 (1) | 0 (0) | 0 (0)
IMPLANT SITE IRRITATION (General disorders) | 0 (0) | 0 (0) | 1 (1)
INFLAMMATION (General disorders) | 2 (2) | 0 (0) | 1 (1)
MALAISE (General disorders) | 1 (1) | 0 (0) | 2 (2)
PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1)
PERFORATED ULCER (General disorders) | 1 (1) | 0 (0) | 0 (0)
PNEUMATOSIS (General disorders) | 1 (1) | 0 (0) | 0 (0)
PRODUCT ADHESION ISSUE (General disorders) | 1 (1) | 0 (0) | 0 (0)
SOFT TISSUE INFLAMMATION (General disorders) | 1 (1) | 0 (0) | 0 (0)
VESSEL PUNCTURE SITE HAEMORRHAGE (General disorders) | 1 (1) | 0 (0) | 1 (1)
XEROSIS (General disorders) | 0 (0) | 0 (0) | 1 (1)
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 76 (81) | 14 (14) | 25 (29)
HEPATIC ENZYME INCREASED (Investigations) | 6 (7) | 13 (13) | 5 (5)
HAEMOGLOBIN DECREASED (Investigations) | 11 (12) | 10 (11) | 7 (11)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 2 (2) | 5 (5) | 4 (4)
OCCULT BLOOD POSITIVE (Investigations) | 3 (3) | 3 (3) | 5 (5)
TRANSAMINASES INCREASED (Investigations) | 4 (4) | 3 (3) | 2 (2)
HAEMATOCRIT DECREASED (Investigations) | 1 (1) | 2 (2) | 1 (1)
OCCULT BLOOD (Investigations) | 2 (2) | 2 (2) | 3 (3)
PROSTATIC SPECIFIC ANTIGEN INCREASED (Investigations) | 1 (1) | 2 (2) | 3 (4)
5-HYDROXYINDOLACETIC ACID INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
BLOOD GLUCOSE ABNORMAL (Investigations) | 0 (0) | 1 (1) | 0 (0)
BLOOD GLUCOSE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
BLOOD POTASSIUM DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
COAGULATION TIME PROLONGED (Investigations) | 1 (1) | 1 (1) | 0 (0)
EJECTION FRACTION ABNORMAL (Investigations) | 1 (1) | 1 (1) | 0 (0)
ELECTROCARDIOGRAM ST SEGMENT DEPRESSION (Investigations) | 0 (0) | 1 (1) | 1 (1)
INTERNATIONAL NORMALISED RATIO DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
SCAN MYOCARDIAL PERFUSION ABNORMAL (Investigations) | 0 (0) | 1 (1) | 0 (0)
WEIGHT DECREASED (Investigations) | 1 (1) | 1 (1) | 0 (0)
ANGIOGRAM (Investigations) | 0 (0) | 0 (0) | 1 (1)
ANTICOAGULATION DRUG LEVEL ABOVE THERAPEUTIC (Investigations) | 1 (1) | 0 (0) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
BLOOD ELECTROLYTES INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
BLOOD OSMOLARITY DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
BLOOD PRESSURE DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
BLOOD PRESSURE INCREASED (Investigations) | 2 (2) | 0 (0) | 2 (2)
BLOOD SODIUM DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
BLOOD UREA INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
CARDIAC OUTPUT DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
CREATININE RENAL CLEARANCE DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
EJECTION FRACTION DECREASED (Investigations) | 2 (2) | 0 (0) | 1 (1)
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 1 (1) | 0 (0) | 2 (2)
HEART RATE DECREASED (Investigations) | 1 (1) | 0 (0) | 2 (2)
HEART RATE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
INTRAOCULAR PRESSURE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
OXYGEN SATURATION DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
PROTHROMBIN TIME PROLONGED (Investigations) | 1 (1) | 0 (0) | 0 (0)
TROPONIN INCREASED (Investigations) | 2 (2) | 0 (0) | 0 (0)
TUMOUR MARKER INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 50 (51) | 47 (47) | 45 (48)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 30 (31) | 37 (37) | 31 (31)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 12 (12) | 20 (20) | 16 (16)
HIP FRACTURE (Injury, poisoning and procedural complications) | 28 (28) | 19 (19) | 29 (29)
RIB FRACTURE (Injury, poisoning and procedural complications) | 15 (15) | 19 (19) | 18 (18)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 10 (10) | 16 (17) | 17 (17)
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 40 (40) | 15 (15) | 16 (16)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 19 (19) | 14 (15) | 12 (14)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 13 (13) | 14 (14) | 13 (13)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 17 (17) | 12 (12) | 19 (19)
LACERATION (Injury, poisoning and procedural complications) | 13 (14) | 12 (12) | 12 (12)
OPERATIVE HAEMORRHAGE (Injury, poisoning and procedural complications) | 10 (11) | 12 (12) | 5 (5)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 40 (43) | 11 (12) | 10 (10)
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 6 (6) | 10 (10) | 7 (7)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 8 (8) | 8 (8) | 5 (5)
TRAUMATIC HAEMORRHAGE (Injury, poisoning and procedural complications) | 9 (9) | 8 (8) | 9 (9)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 8 (8) | 7 (7) | 6 (9)
CONCUSSION (Injury, poisoning and procedural complications) | 10 (10) | 6 (6) | 9 (9)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 7 (8) | 6 (6) | 6 (7)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 7 (7) | 6 (6) | 5 (5)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 5 (5) | 1 (1)
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 4 (4) | 5 (5) | 2 (2)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 4 (4) | 5 (5) | 3 (3)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 13 (13) | 4 (4) | 9 (9)
PUBIS FRACTURE (Injury, poisoning and procedural complications) | 4 (4) | 4 (4) | 9 (9)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 5 (5) | 4 (4) | 1 (1)
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 5 (5) | 3 (3) | 4 (4)
CONTUSION (Injury, poisoning and procedural complications) | 26 (29) | 3 (3) | 15 (15)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 4 (4) | 3 (3) | 6 (6)
FOREARM FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 2 (2)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 1 (1)
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 0 (0)
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 1 (1)
POST PROCEDURAL HAEMATURIA (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 1 (2)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 4 (4)
ULNA FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 1 (1)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 2 (2)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 5 (5) | 3 (3) | 4 (4)
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 6 (6) | 2 (2) | 9 (9)
ACETABULUM FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 1 (1)
ANASTOMOTIC LEAK (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 3 (3)
FRACTURED SACRUM (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1)
HAND FRACTURE (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 1 (1)
HEAD INJURY (Injury, poisoning and procedural complications) | 10 (10) | 2 (2) | 9 (9)
INCISION SITE HAEMATOMA (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 2 (2)
INJURY (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 0 (0)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 7 (7) | 2 (2) | 1 (1)
LIGAMENT INJURY (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
MENISCUS LESION (Injury, poisoning and procedural complications) | 3 (4) | 2 (2) | 4 (5)
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1)
PERIPROSTHETIC FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
POST CONCUSSION SYNDROME (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
SPINAL COLUMN INJURY (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 5 (5)
SUBCUTANEOUS HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 6 (6) | 2 (2) | 3 (3)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 7 (7) | 2 (2) | 6 (6)
WOUND (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 2 (2)
ANAPHYLACTIC TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
AORTIC INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
BLAST INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
BRAIN CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
BURNS FOURTH DEGREE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
CHEMICAL PERITONITIS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 1 (1)
COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
ELECTRIC SHOCK (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
ESCHAR (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
EXCORIATION (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 0 (0)
EYE INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
FOREIGN BODY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
FRACTURE DISPLACEMENT (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
IN-STENT ARTERIAL RESTENOSIS (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (2)
IN-STENT CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 1 (1)
INTESTINAL ANASTOMOSIS COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
JAW FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
JOINT INJURY (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 1 (1)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 1 (1)
MUSCLE INJURY (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
OVERDOSE (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0)
PERIORBITAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
PERIRENAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
PNEUMOTHORAX TRAUMATIC (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
POCKET EROSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
POSTOPERATIVE ILEUS (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
RADIATION PNEUMONITIS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
SCAPULA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
SHUNT MALFUNCTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
SKELETAL INJURY (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
SKIN INJURY (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
SKULL FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1)
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
TRAUMATIC ARTHRITIS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
VASCULAR GRAFT OCCLUSION (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 3 (3)
VASCULAR INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 4 (4)
WOUND EVISCERATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
WOUND HAEMORRHAGE (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0)
ABDOMINAL WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
AFFERENT LOOP SYNDROME (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 1 (1)
ANAESTHETIC COMPLICATION PULMONARY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
ANASTOMOTIC HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
ANASTOMOTIC ULCER (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
ARTERIAL INJURY (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
ARTERIAL RESTENOSIS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
BURNS SECOND DEGREE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
BURNS THIRD DEGREE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
CARBON MONOXIDE POISONING (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
CARDIAC PROCEDURE COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
CARTILAGE INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
CEREBRAL HAEMORRHAGE TRAUMATIC (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
CHEST INJURY (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
EXTRADURAL HAEMATOMA (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
EYEBALL RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
FACE INJURY (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
FRACTURED COCCYX (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
FRACTURED ISCHIUM (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
GALLBLADDER INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
GASTROSTOMY FAILURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
HAEMATURIA TRAUMATIC (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
HEAT ILLNESS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
INCISION SITE HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
INTENTIONAL OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
KIDNEY RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
LIMB CRUSHING INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
LIMB INJURY (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 1 (1)
MUSCLE RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 4 (4)
OPEN WOUND (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
PERIORBITAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
POISONING (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
POST GASTRIC SURGERY SYNDROME (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
POST LAMINECTOMY SYNDROME (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
POST-TRAUMATIC PAIN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
POSTOPERATIVE RESPIRATORY DISTRESS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
POSTPERICARDIOTOMY SYNDROME (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
RADIATION SKIN INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
RENAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
RESPIRATORY FUME INHALATION DISORDER (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
SKULL FRACTURED BASE (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
SOFT TISSUE INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
SPLENIC RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
STERNAL FRACTURE (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 0 (0)
TENDON INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
THERMAL BURN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
TRACHEAL INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
TRAUMATIC INTRACRANIAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
TWIDDLER'S SYNDROME (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
URINARY RETENTION POSTOPERATIVE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
VASCULAR GRAFT COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
WOUND HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
WOUND NECROSIS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
WOUND SECRETION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (2)
AORTIC ANEURYSM REPAIR (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
CARDIAC PACEMAKER REPLACEMENT (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
COLECTOMY (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
HIP ARTHROPLASTY (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
ARTHRODESIS (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
EPIDURAL BLOOD PATCH (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
IMMOBILE (Social circumstances) | 0 (0) | 2 (2) | 0 (0)
ACTIVITIES OF DAILY LIVING IMPAIRED (Social circumstances) | 0 (0) | 0 (0) | 1 (1)
CARDIAC ASSISTANCE DEVICE USER (Social circumstances) | 1 (1) | 0 (0) | 0 (0)
PHYSICAL DISABILITY (Social circumstances) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Warfarin/Placebo Edoxaban (N=7012) | High Dose Edoxaban/Placebo Warfarin (N=7012) | Low Dose Edoxaban/Placebo Warfarin (N=7002)
urinary tract infection (Infections and infestations) | 703 | 688 | 698
nasopharyngitis (Infections and infestations) | 620 | 620 | 645
bronchitis (Infections and infestations) | 572 | 567 | 584
upper respiratory tract infection (Infections and infestations) | 445 | 411 | 443
anaemia (Blood and lymphatic system disorders) | 242 | 368 | 261
dizziness (Nervous system disorders) | 592 | 514 | 537
headache (Nervous system disorders) | 336 | 334 | 356
atrial fibrillation (Cardiac disorders) | 491 | 474 | 528
cardiac failure (Cardiac disorders) | 448 | 425 | 373
hypertension (Vascular disorders) | 438 | 481 | 475
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 470 | 456 | 434
cough (Respiratory, thoracic and mediastinal disorders) | 365 | 383 | 416
diarrhoea (Gastrointestinal disorders) | 499 | 482 | 486
back pain (Musculoskeletal and connective tissue disorders) | 478 | 476 | 496
arthralgia (Musculoskeletal and connective tissue disorders) | 386 | 385 | 417
oedema peripheral (General disorders) | 675 | 577 | 578
fall (Injury, poisoning and procedural complications) | 565 | 453 | 452

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A study site may not publish results of a study until after a coordinated multicenter publication has been submitted for publication or until one year after the study has ended, whichever occurs first. The study site will have the opportunity to publish results of the study, provided Daiichi Sankyo has had the opportunity to review and comment on the study site's proposed publication prior to being submitted for publication with the advice of patent council and need for subject protection.